

### CLINICAL PROTOCOL

A randomized, single blind, single center, single dose, two period, two sequence crossover bioequivalence study of esomeprazole 20 mg delayed-release capsules (Catalent, Guayama) compared to the esomeprazole 20 mg delayed-release capsules (Nexium 24HR] AstraZeneca Södertälje) in healthy adult subjects under fasted conditions

Protocol Number: 218246

Compound/Product Name: Nexium 24HR

**United States (US) Investigational** 

**New Drug (IND) Number:** 

Not applicable

**European Clinical Trials Database** 

(EudraCT) Number:

Not applicable

Other Regulatory Agency Identified

Number:

Health Canada CTA number HC6-024-

c259857

Phase:

This document contains confidentiality statements that are not relevant for this publicly available version



# **Sponsor Information**

| Sponsor Name & Legal<br>Registered Address | GlaxoSmithKline Consumer Healthcare (UK) Trading Limited |
|---|---|
| | 980 Great West Road, |
| | Brentford, |
| | Middlesex, |
| | TW8 9GS, |
| | United Kingdom (UK) |
| Sponsor Contact Details | GlaxoSmithKline Consumer Healthcare (GSK CH) |
| | 184 Liberty Corner Rd., Warren, NJ 07059 United State |

Protocol Number: 218246



# **Document History**

| Document | Version | Summary of Changes |
|---|---|---|
| Original protocol | 1.0 | Not applicable (N/A) |
| | 1.0 | <ul> <li>Page 1: included Health Canada CTA number</li> <li>Table 1-1 Schedule of Activities: Inclusion exclusion criteria check is performed on Day 1 instead of Day -1</li> <li>Exclusion criteria # 22 change for clarification</li> <li>Section 5.5.1 change for clarification</li> <li>Section 5.5.4 change for clarification</li> <li>Table 6.1 Investigational/Study product Supplies Product Master Formulation Code (MFC) corrected</li> <li>Section 6.1 change for clarification</li> <li>Section 7.1 change of text on withdrawal criteria</li> <li>Section 8.2.1: Inclusion exclusion criteria check is</li> </ul> |
| | | <ul> <li>performed on Day 1 instead of Day -1</li> <li>Section 8.2.2: Inclusion exclusion criteria check is performed on Day 1 instead of Day -1</li> <li>Section 8.2.5: Inclusion exclusion criteria check is performed on Day 1 instead of Day -1</li> <li>Section 8.2.6: Inclusion exclusion criteria check is performed on Day 1 instead of Day -1</li> <li>Section 9.3.1: text deleted for consistency with the process</li> <li>Section 12.3.8 corrected text</li> </ul> |

Amendments incorporate all revisions to date, including amendments made at the request of country health authorities, institutional review boards/ethics committees (IRBs/ECs), etc.



## Principal Investigator Protocol Agreement Page

- I confirm agreement to conduct the study in compliance with the protocol and any amendments according to the current International Conference on Harmonisation Good Clinical Practice (ICH GCP) guidelines.
- I acknowledge that I am responsible for overall study conduct. I agree to personally
  conduct or supervise the described study.
- I agree to ensure that all associates, colleagues and employees assisting in the conduct of
  the study are informed about their obligations. Mechanisms are in place to ensure site staff
  receives all appropriate information throughout the study.
- I agree to conduct this study in full conformance with the laws and regulations of the country in which the research is conducted and the Declaration of Helsinki.

| Investigator Name: | PPD |
|------------------------------|-----------------|
| Investigator Qualifications: | B.Sc., MD |
| Investigator Signature: | PPD |
| Date of Signature/Agreement: | PPD DD-Mmm-YYYY |

Protocol Number: 218246



| Ta | ble o | f Contei | nts | |
|---|---|---|---|---|
| | Spon | sor Inforn | nation | 2 |
| | Docu | ıment Hist | tory | 3 |
| | Princ | ipal Inves | stigator Protocol Agreement Page | 4 |
| | Table | e of Conte | ents | 5 |
| 1 | PRO | TOCOL S | SUMMARY | 11 |
| | 1.1 | Synops | is | 11 |
| | 1.2 | Schedu | le of Activities | 14 |
| 2 | INTE | RODUCTI | ION | 16 |
| | 2.1 | Study E | Background and Rationale | 16 |
| | 2.2 | Benefit | /Risk Assessment | 16 |
| | 2.3 | Mechar | nism of Action/Indication | 16 |
| 3 | STU | DY OBJE | CTIVES AND ENDPOINTS | 16 |
| 4 | STU | DY DESI | GN | 18 |
| | 4.1 | Overall | Design | 18 |
| | 4.2 | Scientif | fic Rationale for Study Design | 19 |
| | 4.3 | Justifica | ation for Dose | 19 |
| | 4.4 | End of | Study Definition | 19 |
| 5 | STU | DY POPU | JLATION | 20 |
| | 5.1 | Type ar | nd Planned Number of Subjects | 20 |
| | 5.2 | Inclusio | on Criteria | 20 |
| | 5.3 | Exclusi | on Criteria | 21 |
| | 5.4 | Randon | nization Criteria | 23 |
| | 5.5 | Lifestyl | le Considerations | 23 |
| | | 5.5.1 | Meals and Dietary Restrictions | 23 |
| | | 5.5.2 | Alcohol, Caffeine and Tobacco | 24 |
| | | 5.5.3 | Activity | 24 |
| | | 5.5.4 | Contraception | 24 |
| | 5.6 Screen Failures | | | 25 |
| | 5.7 Sponsor's Qualified Medical Personnel | | | |
| | 5.8 Rater/Clinical Assessor Qualifications | | | |
| 6 | INVI | ESTIGAT | IONAL/STUDY PRODUCTS | 26 |





| | 6.1 | Investig | gational/Study Product Supplies | 26 |
|---|---|---|---|---|
| | | 6.1.1 | Dosage Form and Packaging | 29 |
| | | 6.1.2 | Preparation and Dispensing | 29 |
| | 6.2 | Admini | istration | 29 |
| | | 6.2.1 | Medication/Dosing Errors | 30 |
| | | 6.2.2 | Overdose | 30 |
| | 6.3 | Investig | gational/Study Product Storage | 31 |
| | 6.4 | Investig | gational/Study Product Accountability | 31 |
| | | 6.4.1 | Destruction of Investigational/Study Product Supplies | 32 |
| | 6.5 | Blindin | g and Allocation/Randomization | 32 |
| | 6.6 | Breakir | ng the Blind | 32 |
| | 6.7 | Compli | ance | 33 |
| | 6.8 | Concor | nitant Medication/Treatment(s) | 33 |
| 7 | DISC | SISCONTINUATION OF STUDY INTERVENTION AND SUBJECT | | |
| | DISC | | JATION/WITHDRAWAL | |
| | 7.1 | Subject | t Discontinuation/Withdrawal | 33 |
| | 7.2 | Lost to | Follow up | 34 |
| 8 | STUL | OY PROC | CEDURES | 35 |
| | 8.1 | Visit 1/ | Screening | 35 |
| | | 8.1.1 | Informed Consent | 35 |
| | | 8.1.2 | Demographics | 36 |
| | | 8.1.3 | Inclusion/Exclusion Criteria | 36 |
| | | 8.1.4 | Medical History and Prior Medication/Treatment | 36 |
| | | 8.1.5 | Subject Eligibility | 36 |
| | | 8.1.6 | Screening Procedures | 36 |
| | 8.2 | Study F | Period | 37 |
| | | 8.2.1 | Period 1/Day -1 | 38 |
| | | 8.2.2 | Period 1/Day 1 | 39 |
| | | 8.2.3 | Period 1/Day 2 | 39 |
| | | 8.2.4 | Washout Period | 40 |
| | | 8.2.5 | Period 2/Day -1 | 40 |
| | | 8.2.6 | Period 2/Day 1 | 41 |

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH SOP-208661 Clinical Protocol Template v7.0

## Protocol Number: 218246



| | | 8.2.7 | Period 2/Day 2 | 42 |
|---|---|---|---|---|
| | | 8.2.8 | End of Study | 42 |
| | 8.3 | Study C | onclusion | 42 |
| | 8.4 | Follow- | up Visit | 43 |
| 9 | STUE | Y ASSE | SSMENTS | 43 |
| | 9.1 | Screenin | ng Assessments | 43 |
| | 9.2 | Safety a | and Other Assessments | 43 |
| | | 9.2.1 | Laboratory Tests | 43 |
| | | 9.2.2 | Serology | 45 |
| | | 9.2.3 | Urine drug screen | 45 |
| | | 9.2.4 | Alcohol test | 45 |
| | | 9.2.5 | Pregnancy Testing | 45 |
| | | 9.2.6 | Physical Examinations | 46 |
| | | 9.2.7 | Height and Weight | 46 |
| | | 9.2.8 | Blood Pressure and Pulse Rate | 46 |
| | | 9.2.9 | Respiratory Rate | 47 |
| | | 9.2.10 | Temperature | 47 |
| | | 9.2.11 | COVID-19 Test | 47 |
| | | 9.2.12 | Electrocardiogram | 47 |
| | 9.3 | Pharma | cokinetics (PK) | 48 |
| | | 9.3.1 | Plasma for analysis of esomeprazole | 48 |
| | | 9.3.2 | Shipment of Pharmacokinetic Samples | 48 |
| | 9.4 | Blood V | <sup>7</sup> olume | 49 |
| 10 | ADV | ERSE EV | ENT AND SERIOUS ADVERSE EVENTS | 49 |
| | 10.1 | Definiti | on of an Adverse Event (AE) | 49 |
| | 10.2 | Definiti | on of a Serious Adverse Event (SAE) | 50 |
| | 10.3 | Time Pe | eriod and Frequency for Collecting AE and SAE Information | 52 |
| | 10.4 | Reportin | ng Procedures | 52 |
| | | 10.4.1 | Reporting of an Adverse Event | 53 |
| | | 10.4.2 | Reporting of a Serious Adverse Event | 53 |
| | 10.5 | Evaluati | ing Adverse Events | |
| | | 10.5.1 | Assessment of Intensity | 54 |

Protocol Number: 218246



| | | 10.5.2 | Assessment of Causality | 54 |
|---|---|---|---|---|
| | 10.6 | Follow-u | p of AEs and SAEs | 55 |
| | 10.7 | Withdray | wal Due to an Adverse Event | 56 |
| | 10.8 | Regulato | ry Reporting Requirements for SAEs | 56 |
| | 10.9 | Pregnanc | ey | 57 |
| | | 10.9.1 | Time Period for Collecting Pregnancy Information | 57 |
| | | 10.9.2 | Action to be Taken if Pregnancy Occurs | 57 |
| | 10.10 | Regulato | ry Reporting Requirements for Medical Device Incidents | 57 |
| 11 | DATA | MANAC | GEMENT | 58 |
| | 11.1 | Case Rep | oort Form | 58 |
| | 11.2 | Data Har | ndling | 59 |
| | | 11.2.1 | Data Queries | 59 |
| | 11.3 | External | Data | 59 |
| 12 | STAT | ISTICAL | CONSIDERATIONS AND DATA ANALYSES | 60 |
| | 12.1 | Sample S | Size Determination | 60 |
| | 12.2 | Populatio | ons for Analysis | 60 |
| | 12.3 | Statistica | ıl Analyses | 60 |
| | | 12.3.1 | Primary Analysis(es) | 61 |
| | | 12.3.2 | Secondary Analysis(es) | 62 |
| | | 12.3.3 | Safety Analysis(es) | 62 |
| | | 12.3.4 | Other Analysis(es) | 63 |
| | | 12.3.5 | Exclusion of Data from Analysis | 63 |
| | | 12.3.6 | Demographic and Baseline Characteristics | 63 |
| | | 12.3.7 | Study Drug/Product Compliance and Use of Other Therapies | 63 |
| | | 12.3.8 | Handling of Dropouts and Missing Data | 63 |
| | | 12.3.9 | Interim Analysis | 64 |
| 13 | STUD | Y GOVE | RNANCE CONSIDERATIONS | 64 |
| | 13.1 Quality Control | | | |
| | 13.2 | Quality A | Assurance | 64 |
| | 13.3 | Regulato | ry and Ethical Considerations | 65 |
| | | 13.3.1 | Institutional Review Board/ Ethics Committee | 65 |
| | | 13.3.2 | Ethical Conduct of the Study | 65 |

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH SOP-208661 Clinical Protocol Template v7.0



| | | 13.3.3 | Subject Information and Consent | 66 |
|---|---|---|---|---|
| | | 13.3.4 | Subject Recruitment | 66 |
| | | 13.3.5 | Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 66 |
| | 13.4 | Posting o | f Information on Publicly Available Clinical Trial Registers | 67 |
| | 13.5 | Provision | of Study Results to Investigators | 67 |
| | 13.6 | Records 1 | Retention | 67 |
| | 13.7 | Condition | ns for Terminating the Study | 68 |
| 14 | REFE | RENCES. | | 69 |
| 15 | APPE | NDICIES. | | 70 |
| | 15.1 | ABBREV | VIATIONS | 70 |

Protocol Number: 218246



## List of in text tables

| Table 1-1 | Schedule of Activities | 14 |
|-----------|----------------------------------------|----|
| Table 3-1 | Study Objectives and Endpoints | 16 |
| Table 6-1 | Investigational/Study Product Supplies | 27 |
| Table 6-2 | Sundry Items | 28 |
| Table 9-1 | Laboratory Tests | 44 |
| Table 9-2 | Blood Volume | 49 |



## 1 PROTOCOL SUMMARY

## 1.1 Synopsis

#### **Short Title:**

A bioequivalence study of 20 mg esomeprazole delayed-release capsule (Catalent, Guayama) compared to the current marketed 20 mg esomeprazole delayed-release capsule (Nexium 24HR, AstraZeneca [AZ] Södertälje) in healthy adult subjects under fasting conditions.

## **Background and Rationale:**

This study will be conducted to support the registration of Catalent (Winchester, KY) and Guayama (Puerto Rico) (Encapsulation Only) as alternate sites by determining whether the esomeprazole capsules 20 mg pellets manufactured at Catalent and encapsulated at Guayama (CG) (test product) are bioequivalent to esomeprazole capsules 20 mg from AZ (reference product) under fasted conditions. The data collected will be used for registration and approval for the esomeprazole capsules 20 mg from Catalent and Guayama (Encapsulation Only).

### **Objectives and Endpoints:**

| Objective(s) | Endpoint(s) |
|---|---|
| Primary | |
| Demonstrate the bioequivalence of esomeprazole 20 mg delayed-release capsules from Catalent Guayama (CG) compared to esomeprazole 20 mg delayed-release capsules from AstraZeneca Södertälje (AZ) under fasted conditions | <ul> <li>C<sub>max</sub> (The maximum observed post-dose concentration; obtained without interpolation)</li> <li>AUC<sub>0-t</sub> (The area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule)</li> </ul> |
| Secondary | |
| Pharmacokinetics | |
| Assess the pharmacokinetic profile | <ul> <li>AUC<sub>0-inf</sub> (The area under the plasma concentration versus time curve calculated from time 0 to infinity AUC<sub>0-inf</sub> = AUC<sub>0-t</sub> + C(t)/λ<sub>z</sub> where C(t) is the concentration at the last measurable sampling time point and λ<sub>z</sub> is the terminal elimination rate constant)</li> <li>%AUC<sub>ex</sub> (Percentage of AUC<sub>0-inf</sub> obtained by extrapolation, calculated as (1-[AUC<sub>0-t</sub>/AUC<sub>0-inf</sub>])×100)</li> </ul> |



| | <ul> <li>λ<sub>z</sub> (The terminal elimination rate constant computed as the slope of the regression line of ln (C(t)) on time. The regression should generally involve at least 3 consecutive measurable concentrations that decrease over time)</li> <li>t<sub>max</sub> (The time of the maximum observed post-dose concentration)</li> <li>t<sub>1/2</sub> (The elimination half-life computed as t<sub>1/2</sub> = ln(2)/ λ<sub>z</sub>)</li> </ul> |
|---|---|
| Safety | |
| Assess the safety profile (local and systemic) of both products | <ul> <li>Monitoring and recording of adverse<br/>events</li> </ul> |
| | <ul> <li>Physical examination</li> </ul> |
| | Vital signs |
| | <ul> <li>Laboratory tests</li> </ul> |

## **Study Design:**

This is a single center, single dose, single-blind, randomized, two-sequence, two-period crossover, bioequivalence study in healthy adult subjects with at least a 7-day washout period.

The study is intended to dose in more than one group; all groups will be dosed at the same clinical site and the same protocol requirements and procedures will be followed within each group.

Blood will be sampled regularly at scheduled times for 24 hours following treatment.

Subjects will be randomly assigned to one of 2 treatment sequences and receive a single dose of one of the following treatments in each period following a crossover design:

Treatment A: esomeprazole 20 mg capsules from CG in the fasted state (Test)

Treatment B: esomeprazole 20 mg capsules from AZ in the fasted state (Reference)

The study will consist of an ambulant screening day within 28 days prior to first product administration and two study periods. In each period, subjects will be confined from the day before dosing (Day -1) until 24 hours post-dosing (Day 2), during which pharmacokinetic (PK) blood samples will be obtained within 1 hour prior to dosing (pre-dose) and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, and 24 hours after drug administration. Carry-over effects will be avoided by a wash-out interval of at least 7 days between investigational product administrations.

Following an overnight fast of at least 10 hours, subjects will receive the investigational product in the fasted state with approximately 240 mL of ambient temperature water. Subjects will be instructed to consume the entire amount of water along with their investigational product.



Subjects should swallow the investigational product whole and should not chew or manipulate the medication prior to swallowing.

In order to standardize the conditions on PK sampling days, all subjects should refrain from lying down, eating, and drinking beverages other than water during the first 4 hours after dosing. Aside from time of product administration, water will be allowed *ad libitum* except within 1 hour before and 1 hour after investigational product administration.

For each subject the duration of study participation is 37 days of which up to 2 days confined in each period (total of up to 4 days confined).

## Study Products:

| | Test Product | Reference Product |
|---|---|---|
| Product Name | esomeprazole 20 mg<br>delayed-release capsules | esomeprazole 20 mg<br>delayed-release capsules<br>(Nexium 24HR) (Canadian<br>available product) |
| Dose/Application | One capsule administration | One capsule administration |
| Route of Administration | Oral | Oral |

## Type and Planned Number of Subjects:

A sufficient number of male and female subjects will be screened to randomize approximately 49 to ensure at least 41 evaluable subjects (refer to section 12.1) complete the study.

#### Statistical Methods:

The PK analysis set will be used for the PK evaluations. It includes all subjects of the PK population who complete both treatment periods, and for which the relevant PK parameters (at least AUC<sub>0-t</sub> or C<sub>max</sub>) can be derived. Subjects with baseline concentration >5% of the individual C<sub>max</sub> for either period will be excluded from the PK analysis set. This analysis set will be used in summaries, the primary PK analysis, and the secondary PK analysis.

The PK parameters that will be used in the primary analyses are AUC<sub>0-t</sub> and C<sub>max</sub>.

A linear mixed effects model will be fit to the log-transformed PK parameters (AUC<sub>0-t</sub> and C<sub>max</sub>), as the dependent variable, and treatment, sequence, and period as fixed effects. Subject nested within sequence will be a random effect. The treatment least-squares means (LSMs), difference between treatment LSMs, and 90% confidence interval (CI) for the difference will

Protocol Number: 218246



be computed. The adjusted mean difference and the 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (test/reference) and 90% CIs for the ratio. If all study subjects are not recruited from the same enrollment pool and the study doses in more than one group, the statistical model may be modified to reflect the multigroup nature of the study. Bioequivalence will be declared for AUC<sub>0-t</sub> if the 90% 2-sided CI for the ratio lies completely within the range of 0.8-1.25 and for C<sub>max</sub> if the point estimate for the ratio lies completely within the range of 0.8-1.25. No further adjustments for multiplicity of the co-primary endpoints are necessary as both endpoints must be met in order to achieve study success.

#### 1.2 Schedule of Activities

The schedule of activities table provides an overview of the subject visits and study procedures.

The investigator may schedule visits (unplanned visits) in addition to those listed on the schedule of activities, to conduct evaluations or assessments required to protect the well-being of the subject.

Table 1-1 Schedule of Activities

| Procedure/Assessment | Screening | Treatment Periods 1 and 2ª | | | End of study visit* |
|---|---|---|---|---|---|
| Study day | -28 to -2 | -1 | 1 | 2 | 2 |
| Confinement | | Х | Х | | |
| Discharge | | | | Х | |
| Informed consent | х | | | | |
| Demography | x | | | | |
| Medical history | х | | | | |
| Physical examination <sup>b</sup> | х | Х | | | х |
| Height, weight, BMI | Х | | | | |
| Vital signs (BP, PR, RR, BT) | x | Xc | Xc | Xc | х |
| 12-lead ECG | х | | | | |
| Laboratory tests | х | | | | х |
| COVID-19 test <sup>d</sup> | х | Х | | Х | х |
| Virology | х | | | | |
| Urine pregnancy teste | х | | | | х |
| Serum pregnancy teste | | Х | | | |
| FSH <sup>f</sup> | Х | | | | |
| Urine drug screen | Х | Х | | | |
| Urine cotinine test | х | х | | | |

Protocol Number: 218246



| Procedure/Assessment | Screening | Treatment Periods 1 and 2ª | | | End of study visit* |
|---|---|---|---|---|---|
| Study day | -28 to -2 | -1 | 1 | 2 | 2 |
| Alcohol breath test | х | х | | | |
| Inclusion/exclusion assessment | x | | Xa | | |
| Randomization <sup>h</sup> | | | Х | | |
| Drug administration | | | Х | | |
| PK blood sampling <sup>i</sup> | | | Х | Х | |
| Concomitant treatments | х | х | Х | Х | х |
| Adverse events <sup>j</sup> | х | х | Х | Х | х |

Abbreviations: BMI, BP, PR, RR, BT, ECG, FSH, PK

#### Footnotes:

- \*These assessments are also to be conducted for subjects who discontinue study drug. End of Study visit will occur before discharge, on study Day 2 of Period 2.
- <sup>a</sup>The washout period between each drug administration will be at least 7 days.
- <sup>b</sup>A full physical examination will be performed at screening and a brief physical examination will be performed on Day -1 in each treatment period and end of study.
- <sup>c</sup>Blood pressure (BP), pulse rate (PR), respiratory rate (RR), oral body temperature (BT): pre-treatment on Day 1 (within 1 hour before drug administration) of each treatment period. Oral body temperature (BT) on Day -1 and Day 2 of each treatment period (Note: oral body temperature performed on Day 2 of Period 2 can be used as the oral body temperature required at End of Study).
- <sup>d</sup>Before the first dosing two consecutive tests (locally approved tests [PCR or Antigen]) separated > 24 hours will be performed: one test at screening within 72 hours of admission and one test at check-in (Day-1). Before the second dosing two consecutive tests (locally approved tests [PCR or Antigen]) separated > 24 hours will be performed: one test during the washout period within 72 hours of admission and one test at check-in (Day-1). If the first test is > 72 hours prior to unit admission, subjects should be advised to self -quarantine until entrance to the unit while awaiting final testing clearance. Subjects who report symptoms suggestive of COVID-19 while in the research unit should be isolated in the unit or at home and tested for COVID-19 infection using an approved molecular test. One test (locally approved tests [PCR or Antigen]) should be performed before releasing the subject from the unit in each period or at early discontinuation.
- e for all females of childbearing potential.
- <sup>f</sup>FSH done only in females who have been amenorrhoeic for 12 months
- <sup>9</sup>At the discretion of the Investigator, subjects could continue the study if any deviation to the inclusion/exclusion criteria does not anticipate to alter study integrity.
- hRandomization conducted prior to the first dosing (Period 1).
- PK blood samples will be collected within 1 hour prior to dosing (pre-dose), and at 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, and 24 hours following dosing in each treatment period.

<sup>j</sup>AEs will be collected from time of informed consent.



#### 2 INTRODUCTION

Nexium 24HR, an esomeprazole 20 mg unbanded delayed-release capsule, is approved for non-prescription use in Canada. Esomeprazole 20 mg delayed-release capsules are currently manufactured at AstraZeneca (AZ) in Södertälje, Sweden. GSK CH plans to manufacture esomeprazole 20 mg pellets at Catalent (Winchester, KY). Encapsulation and finished product release will occur at both Catalent (Winchester, KY) and Guayama (Puerto Rico). The sites (Catalent and Guayama) will be registered as alternate to AZ.

## 2.1 Study Background and Rationale

This study will be conducted to support the registration of Catalent and Guayama (Encapsulation Only) as alternate sites by determining whether the esomeprazole capsules 20 mg pellets manufactured at Catalent and capsulated at Guayama (CG) (test product) are bioequivalent to esomeprazole capsules 20 mg from AZ (reference product) under fasted conditions. The data collected will be used for registration and approval for the esomeprazole capsules 20 mg from Catalent and Guayama (Encapsulation Only).

## 2.2 Benefit/Risk Assessment

Complete information for this product may be found in the single reference safety document (SRSD), which for this study is the Nexium 24HR Health Canada Product Monograph (Date of Revision: April 3, 2020).

#### 2.3 Mechanism of Action/Indication

Esomeprazole is the pure S-enantiomer of racemic omeprazole and suppresses gastric acid secretion by specific inhibition of the H+/K+-adenosine triphosphatase enzyme system at the secretory surface of the gastric parietal cell. Because esomeprazole blocks the final step of acid production, this activity leads to inhibition of both basal and stimulated acid secretion. Oral esomeprazole has demonstrated impressive efficacy and safety profiles in the prescription treatment of the following disease states: symptomatic GERD, erosive esophagitis, duodenal ulcers, *Helicobacter pylori*-associated gastric ulcers, risk reduction of non-steroidal anti-inflammatory drug associated peptic ulcers, and hypersecretory conditions, such as Zollinger-Ellison Syndrome. Nexium 24HR is available for self selection over the counter and is indicated for treatment of frequent heartburn for 14 days.

## 3 STUDY OBJECTIVES AND ENDPOINTS

Table 3-1 Study Objectives and Endpoints

| Objective(s) | Endpoint(s) |
|--------------|-------------|
| Primary | |

Protocol Number: 218246



| Demonstrate the bioequivalence of esomeprazole 20 mg delayed-release capsules from Catalent Guayama (CG) compared to esomeprazole 20 mg delayed-release capsules from AstraZeneca Södertälje (AZ) under fasted conditions | <ul> <li>C<sub>max</sub> (The maximum observed post-dose concentration; obtained without interpolation)</li> <li>AUC<sub>0-t</sub> (The area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule)</li> </ul> |
|---|---|
| Secondary | |
| Pharmacokinetics | |
| Assess the pharmacokinetic profile | <ul> <li>AUC<sub>0-inf</sub> (The area under the plasma concentration versus time curve calculated from time 0 to infinity AUC<sub>0-inf</sub> = AUC<sub>0-t</sub> + C(t)/λ<sub>z</sub> where C(t) is the concentration at the last measurable sampling time point and λ<sub>z</sub> is the terminal elimination rate constant)</li> <li>%AUC<sub>ex</sub> (Percentage of AUC<sub>0-inf</sub> obtained by extrapolation, calculated as (1-[AUC<sub>0-t</sub>/AUC<sub>0-inf</sub>])×100)</li> </ul> |
| | <ul> <li>λz (The terminal elimination rate constant computed as the slope of the regression line of ln (C(t)) on time. The regression should generally involve at least 3 consecutive measurable concentrations that decrease over time)</li> <li>t<sub>max</sub> (The time of the maximum observed post-dose concentration)</li> <li>t<sub>1/2</sub> (The elimination half-life computed</li> </ul> |
| Safety | as $t_{1/2} = \ln(2)/\lambda_z$ |
| Assess the safety profile (local and systemic) of both products | <ul> <li>Monitoring and recording of adverse events</li> <li>Physical examination</li> <li>Vital signs</li> <li>Laboratory tests</li> </ul> |

This study will be considered successful if bioequivalence is demonstrated between esomeprazole 20 mg delayed-release capsules from CG and the esomeprazole 20 mg delayed-release capsules from AZ.



#### 4 STUDY DESIGN

## 4.1 Overall Design

This is a single center, single dose, single-blind, randomized, two-sequence, two-period crossover, bioequivalence study in healthy adult subjects with at least a 7-day washout period.

The study is intended to dose in more than one group; all groups will be dosed at the same clinical site and the same protocol requirements and procedures will be followed within each group.

Blood will be sampled regularly at scheduled times for 24 hours following treatment.

Subjects will be randomly assigned to one of 2 treatment sequences and receive a single dose of one of the following treatments in each period following a crossover design:

Treatment A: esomeprazole 20 mg capsules from CG in the fasted state (Test)

Treatment B: esomeprazole 20 mg capsules from AZ in the fasted state (Reference)

The study will consist of an ambulant screening day within 28 days prior to first product administration and two study periods. In each period, subjects will be confined from the day before dosing (Day -1) until 24 hours post-dosing (Day 2), during which time pharmacokinetic (PK) blood samples will be obtained within 1 hour prior to dosing (pre-dose) and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, and 24 hours after drug administration. Carry-over effects will be avoided by a wash-out interval of at least 7 days between investigational product administrations.

Following an overnight fast of at least 10 hours, subjects will receive the investigational product in the fasted state with approximately 240 mL of ambient temperature water. Subjects will be instructed to consume the entire amount of water along with their investigational product. Subjects should swallow the investigational product whole and should not chew or manipulate the medication prior to swallowing.

In order to standardize the conditions on PK sampling days, all subjects should refrain from lying down, eating, and drinking beverages other than water during the first 4 hours after dosing. Aside from time of product administration, water will be allowed *ad libitum* except within 1 hour before and 1 hour after investigational product administration.

For each subject the duration of study participation is 37 days of which up to 2 days confined in each period (total of up to 4 days confined).

Figure 4-1 Study design

| Screening | Period 1 and 2 <sup>a</sup> | End of study |
|---------------|-----------------------------|-------------------|
| Day -28 to -2 | Day -1 to 2 | Day 2 of Period 2 |

<sup>&</sup>lt;sup>a</sup> Washout period of at least 7 days between each dosing



A sufficient number of male and female subjects will be screened to randomize approximately 49 to ensure at least 41 evaluable subjects (refer to section 12.1) complete the entire study.

## 4.2 Scientific Rationale for Study Design

Blinding is required as per Canadian regulation. This will be a single-blind study.

Subject will be blinded to treatment; test and reference product are identical.

The degree of blinding will depend on the assessment as follows:

- Personnel performing the bioanalytical analysis will be blinded to the randomized treatment.
- Personnel involved in the collection, monitoring, revision, or evaluation of AEs will be blinded to the randomization.
- Personnel who could have an impact on the outcome of the study will be blinded to the randomization.
- Designated pharmacy personnel at the clinical site not directly involved with the clinical aspects of the trial will prepare and dispense the study medication and will be aware of the randomization code.

A crossover design, using the same subjects to test each product, will be used to reduce variability.

The blood sampling times have been chosen based on the information available particularly on esomeprazole absorption, as well as its elimination.

Non smokers have been chosen as the population for this study to reduce variability.

The following guidance have been followed for designing the study:

- Guidance document, Comparative Bioavailability Standards: Formulations Used for System Effects (Health Canada 2018)
- Guidance document, Conduct and Analysis of Comparative Bioavailability Studies (Health Canada 2018)

#### 4.3 Justification for Dose

This is a study to assess the bioequivalence of the test product to a commercial reference product.

## 4.4 End of Study Definition

A subject is considered to have completed the study if he or she has completed all phases of the study including the last visit or the last scheduled procedure shown in the Schedule of Activities.



The end of this study is defined as the date of the last visit of the last subject to complete the study.

#### 5 STUDY POPULATION

## 5.1 Type and Planned Number of Subjects

A sufficient number of male and female subjects will be screened to randomize approximately 49 to ensure at least 41 evaluable subjects (refer to section 12.1) complete the entire study.

An enrolled subject is one who has agreed to participate in the clinical study following completion of the informed consent process directly and successfully met eligibility criteria to proceed beyond the screening visit as applicable for the protocol design.

This study can fulfill its objectives only if appropriate subjects are enrolled. The following eligibility criteria are designed to select subjects for whom participation in the study is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether a subject is suitable for this protocol.

Subject eligibility to participate in the clinical study should be reviewed and documented by an appropriate member of the investigator's study team before subjects are included in the study.

### 5.2 Inclusion Criteria

An individual must meet all the following inclusion criteria to be eligible to be included into the study:

- 1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study before any assessment is performed.
- 2. Male or female subject who, at the time of screening, is between the ages of 18 and 55 years, inclusive.
- 3. Subject who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
- 4. Healthy subject, which is defined as in general good physical health, as judged by the investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
- 5. Body Mass Index (BMI) of 18.5 to 30.0 kg/m<sup>2</sup>; and a total body weight  $\geq$ 50.0 kg for males and  $\geq$ 45.0 kg for females.
- 6. Subject with two negative tests (one at screening within 72 hours of admission and one at check on Day-1) for active COVID-19, separated by > 24 hours.



7. Female subject of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. Female subjects who are not of childbearing potential must meet requirements in the Contraception section of protocol.

#### 5.3 Exclusion Criteria

A subject with any of the following characteristics/conditions will not be included in the study:

- 1. Subject who is an investigational site staff member directly involved in the conduct of the study and his/her family members, site staff member otherwise supervised by the investigator, or subject who is a GSK employee directly involved in the conduct of the study.
- 2. Participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation.
- 3. Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
- 4. Pregnant female subject.
- 5. Breastfeeding female subject.
- 6. Known or suspected intolerance or hypersensitivity or photosensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
- 7. Diagnosis of long QT syndrome or QTc > 450 msec for males and > 470 msec for females at screening.
- 8. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or pulse rate less than 50 or over 100 bpm).
- 9. A subject unwilling or unable to comply with Lifestyle Considerations described in this protocol.
- 10. Use of any medication (including over-the-counter medications and herbal remedies) within 2 weeks before first scheduled study drug administration or within less than 10 times the elimination half-life of the respective drug (whichever is longer), or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:
  - systemic contraceptives and hormone replacement therapy, as long as female subject is on stable treatment for at least 3 months before first scheduled study drug administration and continues treatment throughout the study;
  - occasional use of acetaminophen (up to 2 g daily).



- 11. Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
- 12. Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
- 13. Subject with signs and symptoms suggestive of COVID-19 (i.e. fever, cough, etc)\* within 14 days of inpatient admission. \*as defined by WHO or local guidance)
- 14. Subject with known COVID-19 positive contacts in the past 14 days.
- 15. Any vaccination, including COVID-19 vaccine, within 14 days prior to the first dose.
- 16. Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance but not limited to any of the following:
  - History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, *e.g.*, appendectomy and herniorrhaphy);
  - History of inflammatory bowel disease;
  - History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (> 123 μmol/L for males and > 95 μmol/L for females) or BUN (≥ 12.0 mmol/L) or the presence of clinically significant abnormal urinary constituents (e.g. albuminuria);
  - History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found: 1) AST (≥ 1.2 ULN), ALT (≥ 1.2 ULN), 2) GGT (≥ 1.2 ULN), ALP (≥ 1.2 ULN), 3) bilirubin (≥ 48 µmol/L for males and ≥ 30 µmol/L for females) or CK (≥ 3 ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the investigator;
  - Evidence of urinary obstruction or difficulty in voiding at screening;
  - History or clinical evidence at screening of pancreatic injury or pancreatitis.
- 17. Subject has a history of drug abuse or investigator has evidence of current drug abuse with drug classes that include but are not limited to barbiturates, tricyclic antidepressants, amphetamines, benzodiazepines, cocaine, opiates, cannabis or any other drugs (verified by urine drug screen or other reliable evidence).
- 18. Evidence, as reported by an alcohol breath testing, for current alcohol abuse or reports a regular average alcohol consumption exceeding 18 g (women) or 35 g (men) of pure alcohol per day, i.e. 1 drink/day for women or 2 drinks/day for men (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.

Protocol Number: 218246



- 19. Subject reported regular consumption of > 5 cups of coffee or tea per day (or equivalent consumption of  $\ge 500$  mg xanthine per day using other products)
- 20. Smoker, defined as the use of tobacco or nicotine products during the 3 months prior to screening until admission to the unit or a positive urine cotinine test at screening.
- 21. A subject who is unwilling to abstain from tobacco or nicotine-containing product use during the study.
- 22. Subject reports consumption of any drug metabolizing enzyme (e.g. CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (*e.g.* broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort *etc.*) within 2 weeks prior to admission to the unit.
- 23. Positive results in any of the virology tests for HIV antigen and antibody, HCV Ab, HbsAg, and HBcAb (IgG + IgM).
- 24. Performance of unaccustomed strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission and throughout the entire study.
- 25. Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the investigator's opinion may pose a risk to the candidate.
- 26. Any condition not identified in the protocol that in the opinion of the investigator would confound the evaluation and interpretation of the study data or may put the subject at risk
- 27. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dose.
- 28. Subject who has previously been enrolled in this study.

#### 5.4 Randomization Criteria

Subjects will be randomized into the study provided they have satisfied all subject selection criteria.

## 5.5 Lifestyle Considerations

## 5.5.1 Meals and Dietary Restrictions

- Subjects must abstain from all food and drink (except water) at least 4 hours prior to any safety laboratory evaluations and 10 hours prior to investigational product administration. Water is permitted until 1 hour prior to investigational product administration.
- Water may be consumed without restriction beginning 1 hour after dosing.
- Non-caffeinated drinks (except grapefruit or grapefruit-related citrus fruit juices see below) may be consumed with meals and the evening snack.



- Lunch will be provided approximately 4 hours after dosing.
- Dinner will be provided approximately 12 hours after dosing.
- An evening snack may be permitted approximately 2 hours after evening meal.
- Subjects will not be allowed to eat or drink grapefruit or grapefruit-related citrus fruits (e.g. Seville oranges, pomelos, papaw, dragon fruit, kiwi fruit, mango, passion fruit, pomegranate, rambutan, star fruit or products that contain these fruits) from 2 weeks prior to admission to the unit until collection of the final pharmacokinetic blood sample.
- Meals intake during the study will also be standardized.

#### 5.5.2 Alcohol, Caffeine and Tobacco

- Subjects will abstain from alcohol for 48 hours prior to admission to the clinical site
  in each period and continue abstaining from alcohol until collection of the final
  pharmacokinetic sample of each study period. Subjects will undergo an alcohol breath
  test at screening, at admission to each treatment period and at the discretion of the
  investigator.
- Subjects will abstain from caffeine-containing products for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample of each study period.
- Subjects will abstain from the use of tobacco- or nicotine-containing products including nicotine patches and other delivery devices such as electronic cigarettes or vaporizers) from screening and throughout the study.

## 5.5.3 Activity

- Subjects will not be permitted to assume a fully recumbent position for 4 hours following dosing.
- Subjects will abstain from strenuous exercise (e.g. heavy lifting, weight training, calisthenics, aerobics) for the duration of the study. Walking at a normal pace will be permitted.
- Subjects will abstain from strenuous exercise (e.g., heavy lifting, weight training, calisthenics, aerobics) for at least 48 hours prior to each blood collection for clinical laboratory tests and throughout the entire study. Walking at a normal pace will be permitted.

## 5.5.4 Contraception

All female subjects who are of childbearing potential and are sexually active and at risk for pregnancy must agree to use a highly effective method of contraception consistently and correctly for the duration of the active study period and for 30 days after the last dose of investigational product. The investigator or his or her designee, in consultation with the subject,



will confirm that the subject has selected an appropriate method of contraception for the individual subject from the permitted list of contraception methods (see below) and instruct the subject in its consistent and correct use. Subjects need to affirm that they meet the criteria for the correct use of at least 1 of the selected methods of contraception. The investigator or his or her designee will discuss with the subject the need to use highly effective contraception consistently and correctly according to the schedule of activities and document such conversation in the subject's chart. In addition, the investigator or his or her designee will instruct the subject to call immediately if the selected contraception method is discontinued.

Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (i.e., perfect use) and include the following:

- 1. Established use of oral, inserted, injected, transdermal, or implanted hormonal methods of contraception is allowed provided the subject plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness as deemed appropriate by the investigator;
- 2. Intrauterine contraceptive device (IUD);
- 3. Male condom or female condom used WITH a spermicide (i.e., foam, gel, film, cream, or suppository);
- 4. Male sterilization with absence of sperm in the post-vasectomy ejaculate;
- 5. Bilateral tubal ligation / bilateral salpingectomy or bilateral tubal occlusive procedure (provided that occlusion has been confirmed in accordance with the device's label);
- 6. Female who meets the criteria for non-childbearing potential as described below:

Female subjects of non-childbearing potential must meet at least one of the following criteria:

- Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level ≥40 mIU/mL;
- Have undergone a documented (included self-reported) hysterectomy and/or bilateral oophorectomy.

All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential.

#### 5.6 Screen Failures

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently randomized. To ensure transparent reporting of screen failure subjects, a minimal set of screen failure information will include demography, screen failure details (e.g.



withdrawal of consent), eligibility criteria, any protocol deviations and any adverse events or incidents as applicable.

Individuals who do not meet the criteria for participation in this study (screen failure) may not be re-screened.

## 5.7 Sponsor's Qualified Medical Personnel

Contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the Study Contact List located in the investigator study master file held at the study site.

The contact number is only to be used by investigational staff seeking advice on medical questions or problems in the event that the established communication pathways between the investigational site and the study team are not available.

The contact number is not intended for direct use by study subjects. To facilitate access to appropriately qualified medical personnel on study-related medical questions or problems, subjects will be provided with a contact card. The contact card will provide, as a minimum, protocol identifiers, the subject's study identification number, contact information for the investigational site, and contact details in the event that the investigational site cannot be reached to provide advice on a medical question or problem identified by a healthcare professional other than the investigator.

#### 5.8 Rater/Clinical Assessor Qualifications

No rater/clinical assessor qualifications are required for this study.

#### 6 INVESTIGATIONAL/STUDY PRODUCTS

For the purposes of this study, per International Conference on Harmonization (ICH) guidelines, and GSK policy, study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

This includes a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use.

## 6.1 Investigational/Study Product Supplies

The selection of the Reference product (the currently marketed and commercially available esomeprazole 20 mg capsules from AZ), will be based on assay content to ensure that this product does not differ by more than 5% from that of the batch used as Test product (esomeprazole 20 mg capsules from CG).

Protocol Number: 218246



The following study products will be supplied by the Clinical Supplies Department, GSK CH:

Table 6-1 Investigational/Study Product Supplies

| Table 6-1 Investigational/study Product Supplies | | |
|---|---|---|
| | Test Product | Reference Product |
| Product Name | esomeprazole 20 mg<br>delayed-release capsules | esomeprazole 20 mg<br>delayed-release capsules<br>(Nexium 24HR) (Canadian<br>available product) |
| Pack Design | bottles | bottles |
| Dispensing Details | one capsule once daily | one capsule once daily |
| Product Master Formulation Code (MFC) | CCI | CCI |
| Dose/Application | One capsule administration | One capsule administration |
| Route of Administration | Oral | Oral |
| Usage Instructions | Administer study medication with 240 mL of ambient temperature water Instruct subjects to consume the entire amount of water along with their investigational product | Administer study medication with 240 mL of ambient temperature water Instruct subjects to consume the entire amount of water along with their investigational product |
| Return Requirements | All unused samples to be returned | All unused samples to be returned |

Protocol Number: 218246



## Table 6-2 Sundry Items

Sundry items to be supplied:

| ltem | | Pack<br>Design | Dispensing | Return/Disposal Details | |
|---|---|---|---|---|---|
| | | | Details | Used Samples | Unused<br>Samples |
| Acon 10 Drugs Split<br>Cup | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| BD Vacutainer®,<br>Urine Collection<br>Tubes and Kits, BD<br>Medical | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| Clearview hCG<br>Combo -Pregnancy<br>Tests | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| COT One Step<br>Cotinine Test Device | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| Microtube 2mL PP<br>Jupé, Sans<br>Bouchons | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep at site |
| Tube BD Plastique<br>EDTA K <sub>2</sub> 3mL<br>Lavande | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| Tube BD Plastique<br>SST 3.5mL | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| Tube BD plastique<br>5mL SST | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| Urine Collection Cup<br>with Integrated<br>Transfer Device | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep<br>at site |
| Urine Collection<br>Tube Plastic 8mL | Site/CRO | Commercial pack | Use as per study schedule | Discard/destroy at site using site disposal procedures | To keep at site |
| Regular Polyester<br>Swab with Plastic<br>Applicator | Biomedical<br>Laboratory | Commercial pack | Use as per<br>study schedule | Discard/destroy at biomedical laboratory facility using biomedical laboratory disposal procedures | To keep<br>at site |



Equivalent items can also be used based on supplier availability. Detailed instructions for the return of study product/study supplies for the accountability checks and subsequent destruction which will be provided by GSK CH during the study in time for study close out visit. Sundry items will be supplied by the site/vendor and will be discarded or destroyed at the clinical site.

### 6.1.1 Dosage Form and Packaging

Capsules will be supplied to the clinical site as packaged bottles for dispensing by the pharmacy.

The content of the product labels will be in accordance with all applicable regulatory requirements and will be the responsibility of the GSK CH Global Clinical Supplies group. Each study label will contain, but not be limited to, protocol number, directions for use and storage requirements.

Care should be taken with the supplied products and their labels so that they are maintained in good condition. It is important that all labels remain intact and legible for the duration of the study. Subjects should be instructed to not remove or deface any part of the study label.

All products supplied are for use only in this clinical study and should not be used for any other purpose.

#### 6.1.2 Preparation and Dispensing

Subjects will be assigned to products in accordance with the randomization schedule generated by PPD , prior to the start of the study, using validated software.

Esomerazole capsules will be dispensed by qualified site personnel (unblinded) per the dosage/administration instructions. These staff members will not be involved in any safety, efficacy assessments or other aspects of the study that could be influenced by the knowledge of which product a subject has been assigned to use. An additional member of site staff should ensure the dispensing procedures are completed accurately.

#### 6.2 Administration

Only subjects enrolled in the study may receive study products and only authorized site staff may supply or administer study products. All study interventions must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the authorized site staff only.

Following an overnight fast of least 10 hours, subjects will receive investigational product. Investigator site personnel will administer investigational product during each period with ambient temperature water to a total volume of 240 mL and will instruct subjects to consume the entire amount of water along with their investigational product. A hand and mouth check will be performed to ensure consumption of the medication.



Subjects will swallow the investigational product whole and will not manipulate or chew the medication prior to swallowing. To standardize the conditions on pharmacokinetic sampling days, all subjects will be required to refrain from lying down (except when required by procedures), eating, and drinking beverages for the first 4 hours after dosing. Water may be given after 1 hour post-dosing.

### 6.2.1 Medication/Dosing Errors

Medication/dosing errors may result, in this study, from the administration or consumption of:

- the wrong product,
- by the wrong subject,
- at the wrong time,
- or at the wrong dosage.

Such medication/dosing errors occurring to a study subject are to be captured in the CRF. In the event of medication dosing error, the sponsor should be notified **immediately and under no circumstance should this exceed 24 hours.** 

Medication/dosing errors are reportable irrespective of the presence of an associated AE, including:

- Medication/dosing errors involving subject exposure to any of the study products;
- Potential medication/dosing errors or uses outside of what is foreseen in the protocol that do or do not involve the participating subject.

If a medication/dosing error is accompanied by an AE, as determined by the investigator, the medication/dosing error and, any associated adverse event(s) are to be captured in the CRF AE form.

#### 6.2.2 Overdose

An overdose is a deliberate or inadvertent administration of a product at an amount higher than specified in the protocol.

Overdose is not likely to occur in this study.

Overdose per se is not an AE. However, any clinical sequelae of an overdose should be reported as an AE (and serious adverse event (SAE), if appropriate). For reporting, follow the AE and SAE reporting instructions.



## 6.3 Investigational/Study Product Storage

The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study products received and any discrepancies are reported and resolved before use according to the supplied shipping documentation.

The investigator, or designee, will ensure that all study products are stored in a secured area with controlled access under required storage conditions and in accordance with applicable regulatory requirements and the product label.

Site systems must be capable of measuring and documenting (for example, via a log), at a minimum, daily minimum and maximum temperatures for all site storage locations (as applicable, including frozen, refrigerated, and/or room-temperature products). This should be captured from the time of first product receipt throughout the study. Even for continuous monitoring systems, a log or site procedure that ensures active daily evaluation for excursions should be available. The operation of the temperature-monitoring device and storage unit (for example, refrigerator), as applicable, should be regularly inspected to ensure it is maintained in working order.

Any excursions from the product-label storage conditions should be reported to appropriate site staff upon discovery and communicated to sponsor as soon as possible. The site should actively pursue options for returning the product to the storage conditions as described in the labeling, as soon as possible. Excursions from the storage requirements, including any actions taken, must be documented as a protocol deviation and reported to the Sponsor.

Once an excursion is identified, the affected product (or products) must be quarantined and not used until the sponsor provides documentation of permission to use. Use of any of the affected product(s) prior to sponsor approval will be considered a protocol deviation.

## 6.4 Investigational/Study Product Accountability

All products supplied are for use only in this clinical study and should not be used for any other purpose.

All study products must be received by a designated person at the study sites, handled and stored safely and properly, and kept in a secured location to which only the staff have access. Upon receipt, all study products should be stored according to the instructions specified on the product labels. Study products are to be dispensed only to subjects enrolled in the study in accordance with the protocol, by authorized site staff.

The investigative site must maintain adequate records documenting the receipt, use, loss, or other disposition of all the product supplies. All study products will be accounted for using the investigational/study product accountability form/record. The investigator is responsible for study product accountability, reconciliation, and record maintenance.



The accountability records must be available for inspection by the study monitor during the study. Monitoring of product accountability will be performed by the monitor during site visits and at the completion of the study.

## 6.4.1 Destruction of Investigational/Study Product Supplies

At the end of the study, the investigator or an appropriate designee, and a representative of GSK CH (study monitor) will inventory all used and unused study products and sundry items. The investigational/study product accountability record for returned study products will then be completed. All study product (used and unused) for this clinical study (including empty packaging bottles), will be returned for destruction to the GSK CH Clinical Supplies Department or designated vendor using the return instructions provided. Detailed instructions for the return of study product/study supplies for the accountability checks and subsequent destruction will be provided by GSK CH during the study in time for study close out visit.

## 6.5 Blinding and Allocation/Randomization

The investigator's knowledge of the treatment should not influence the decision to enroll a particular subject or affect the order in which subjects are enrolled.

will provide a randomization schedule to the investigator and, in accordance with the randomization numbers, the subject will receive the study treatment regimen assigned to the corresponding randomization number.

Treatments will be provided in a blind manner. Personnel involved in the collection, monitoring, revision, or evaluation of adverse events, personnel of the bioanalytical department, and personnel who could have an impact on the outcome of the study, including GSK/PPD statisticians, programmers, scientists, DM study managers, clinical study team except Global supply, and PPD PK analyst, will not have prior access to the randomization code.

## 6.6 Breaking the Blind

A paper copy of the randomization list will be kept by the PPD research pharmacy group in a paper envelope, which itself will be inserted in a plastic envelope closed with a secure seal with the medication documents, in a secure place with controlled access, throughout the study. The plastic envelope will be identified in a window, with at least the type of content and the project number. A form will also be provided for documenting the opening and closing of the plastic envelope at PPD . Moreover, the electronic version of the lists will be kept at PPD on a controlled access directory. After the end of study and following PPD project manager's authorization, the randomization list will be opened and kept in the medication binder.



## 6.7 Compliance

Study products will be administered under the supervision of investigator site personnel. A hand and mouth check will be performed to ensure consumption of the medication.

## 6.8 Concomitant Medication/Treatment(s)

Subjects will abstain from all concomitant treatments, except for contraceptives and hormone replacement therapy, and those used for the treatment of adverse events unless they jeopardize the integrity of the study. The study Sponsor should be immediately informed. Any medications, treatments or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) taken during the study, from signing the informed consent, must be recorded in the CRF with indication, reason for use, unit dose, daily dose, and start and stop dates of administration. All subjects will be questioned about medications/treatments at each site visit.

Medication/treatments taken within 90 days of signing the informed consent form will be documented as a prior medication/treatment. Medications/treatments taken after the first dose will be documented as concomitant medication/treatments.

# 7 DISCONTINUATION OF STUDY INTERVENTION AND SUBJECT DISCONTINUATION/WITHDRAWAL

# 7.1 Subject Discontinuation/Withdrawal

A subject may withdraw from the study at any time at his or her own request or may be withdrawn at any time at the discretion of the investigator or sponsor for safety, behavioral reasons, events such as vomiting and diarrhoea which could render the plasma concentration-time profile unreliable or the inability of the subject to comply with the protocol-required schedule of study visits or procedures.

The following circumstances require discontinuation of study product and/or premature subject withdrawal:

- Protocol violation that may impact the subject's safety
- Positive test for COVID-19, conducted during the study, at times deemed necessary by investigator
- Withdrawal of informed consent
- Subject lost to follow-up
- Unblinding of the subject
- Pregnancy



If a subject is discontinued or prematurely withdraws from the study, the reason(s) for discontinuation or withdrawal and the associated date must be documented in the relevant section(s) of the CRF.

## 7.2 Lost to Follow up

If a subject fails to return to the site for a required study visit the site must attempt to contact the subject and reschedule the missed visit as soon as possible and counsel the subject on the importance of maintaining the assigned visit schedule and ascertain whether the subject wishes to and/or should continue in the study.

A subject will be considered lost to follow up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. Before a subject is deemed lost to follow up, the investigator or designee must make every effort to regain contact with the subject (where possible, 3 telephone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods). These contact attempts should be documented. If contact is made with the subject, the investigator should inquire about the reason for withdrawal, request that the subject return all products that they had been dispensed and if appropriate request that the subject return for a final visit and follow-up with the subject regarding any unresolved adverse events (AEs).

Final safety assessments may be carried out when the subject returns to the study site, at the investigator's discretion, which could include the following:

- urine pregnancy test,
- physical examination,
- safety laboratory tests,
- seated blood pressure, respiratory rate, oral body temperature and pulse rate measurements.

Should the subject continue to be unreachable, he/she will be considered to have withdrawn from the study and lost to follow up.

Lack of completion of all or any of the early termination procedures will not be viewed as protocol deviations so long as the subject's safety was preserved.

If the subject withdraws from the study and withdraws consent for disclosure of future information, no further evaluations should be performed, and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.



#### 8 STUDY PROCEDURES

This section lists the procedures to be completed at each planned study visit. The timing of each procedure is listed in the Schedule of Activities section.

Adherence to the study design requirements, including all procedures are essential and required for study conduct.

## 8.1 Visit 1/Screening

Screening procedures will be conducted by the investigator, or suitably qualified designee.

Subjects will be screened within 28 days prior to administration of the investigational product to confirm that they meet the subject selection criteria for the study.

The following procedures will be completed:

#### 8.1.1 Informed Consent

The investigator, or designee, must obtain informed consent from each subject participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study. The informed consent form (ICF) will be signed and dated by the subject. A copy will be given to the subject, and the original signed and dated ICF will be maintained in the subject's records.

The investigator, or designee, must also explain to the subjects that they are completely free to refuse to enter the study or to withdraw from it at any time. Appropriate forms for documenting a signed and dated consent will be provided by either the investigator or by GSK CH.

The investigator, or designee, should sign and date the ICF to confirm that the consent process was completed correctly after the subject has signed.

The time the subject signed the informed consent form will be captured as this is the point at which all adverse events will be captured from. The date and time of consent will be captured in the CRF.

If, during a subject's participation in the study, any new information becomes available that may affect the subject's willingness to participate in the study, each ongoing subject should receive a copy of this new information and be re-consented into the study. Each subject should be provided with a copy of the signed and dated amended consent form. The date of re-consent will be recorded on the CRF.

After signing the ICF, subjects will undergo the screening assessments to confirm that they meet all the inclusion criteria and none of the exclusion criteria. If the subject is confirmed eligible by the investigator (or designee) to participate in the study the subject is considered enrolled in the study.



### 8.1.2 Demographics

The following demographic information will be recorded in the CRF: year of birth, gender, ethnicity and race.

Ethnicity and race of subjects will be recorded in accordance with FDA Guidance for Industry: Collection of Race and Ethnicity Data in Clinical Trials, 2005.

#### 8.1.3 Inclusion/Exclusion Criteria

Inclusion and exclusion criteria information, as specified in Section 5, will be documented in the CRF.

## 8.1.4 Medical History and Prior Medication/Treatment

Details of relevant medical and surgical history (in the last 5 years), including allergies or drug sensitivity, will be documented in the CRF.

Prior medications/treatments, including prescription and non-prescription drugs, dietary supplements and herbal remedies, taken in the last 90 days and prior to signing the informed consent form, will be documented in the CRF.

## 8.1.5 Subject Eligibility

The investigator and/or medically qualified designee will review inclusion/exclusion criteria, medical history, prior medications to confirm subject eligibility to participate in the clinical trial. This will be documented in the CRF.

To prepare for study participation, subjects will be instructed on the Lifestyle Considerations and any Concomitant Medication/Treatment(s) requirements of the protocol.

#### 8.1.6 Screening Procedures

The following procedures will be completed:

- Obtain written informed consent and record in the CRF.
- Review Inclusion and Exclusion criteria and record in the CRF.
- Collect demography, including year of birth, gender, ethnicity and race and record in the CRF.
- Collect height and weight and calculate BMI. The results for each measurement will be recorded in the CRF.
- Obtain medical history as related to the inclusion/exclusion criteria, including any relevant medical or surgical history, allergies or drug sensitivity, history of drug and


alcohol use. Significant findings that are present before consent must be included in the CRF.

- Obtain complete medication history of all prescription or nonprescription drugs, and dietary and herbal supplements taken within 90 days prior to consent, and record in the CRF.
- Obtain seated blood pressure, pulse rate, respiratory rate and oral body temperature. The results for each measurement will be recorded in the CRF.
- Conduct full physical examination. Any clinically relevant findings will be noted in the AE CRF page and enrollment will be based upon investigator judgement.
- Contraceptive review.
- Collect single 12 lead ECG. Results (normal or abnormal) and clinical significance will be recorded on the CRF.
- Following at least a 4 hour fast, collect blood and urine specimens for the following, and recorded on the CRF:
  - Safety laboratory tests and virology;
  - Urine drug screening;
  - Alcohol screening;
  - Cotinine screening;
  - Serum FSH concentration for any female who has been amenorrheic for at least 12 consecutive months;
  - Urine pregnancy test for all females of childbearing potential.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.
- Collect nasal/nasopharyngeal swab sample for COVID-19 test within 24 to 72 hours prior to check-in (Day -1) in Period 1. Date and time of sample collection and test results (positive or negative) will be documented in the CRF.

## 8.2 Study Period

For the study periods described below, when multiple procedures are scheduled at the same time point(s) relative to dosing, the following chronology of events should be adhered to, where possible.



- Blood pressure/pulse rate: obtain as close as possible to scheduled time, but prior to blood specimen collection;
- Pharmacokinetic blood specimens: obtain at scheduled time.

Obtain all other procedures as close as possible to the scheduled time but may be obtained before or after blood.

## 8.2.1 Period 1/Day -1

Subjects will be admitted to the clinical site the day prior to Day 1 dosing.

The following procedures will be completed following admission to the clinical site:

- Obtain oral body temperature. The results for each measurement will be recorded in the CRF.
- Brief physical examination including evaluation of general appearance, heart, lung. The results will be recorded in the CRF.
- Collect urine for drug screening. The results will be recorded in the CRF.
- Collect urine for cotinine screening. The results will be recorded in the CRF.
- Obtain blood for serum  $\beta$  -hCG for all females of childbearing potential. The results will be recorded in the CRF (note: blood for serum  $\beta$  -hCG can be obtained at admission or in the morning of Day -1).
- Collect nasal/nasopharyngeal swab sample for COVID-19 test. Date and time of sample collection and test results (positive or negative) will be documented in the CRF.
- Confirm proper contraception is being used and the results will be recorded on the CRF.
- Collect alcohol breath test. Result will be recorded on the CRF.
- Meals as required in section 5.5.1. Time and consumption of meals will be recorded on CRF.
- Subjects will begin fasting at least 10 hours prior to dosing on Day 1.
- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.

Protocol Number: 218246



## 8.2.2 Period 1/Day 1

**Prior to** dosing, within 1 hour of study drug administration, the following procedures will be completed:

- Obtain seated blood pressure, pulse rate, respiratory rate and oral body temperature. The results for each measurement will be recorded in the CRF.
- Review Inclusion and Exclusion criteria and record in the CRF.
- Randomization.
- Collect a blood sample for pharmacokinetic analysis. Time of blood sampling will be recorded in the CRF.
- After all pre-dose procedures have been completed, administer the investigational product (see Investigational/Study Products section) and record in the CRF.

**After dosing**, the following procedures will be completed:

- Collect blood samples for pharmacokinetic analysis at the following time points after dosing on Day 1: 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, and 16 hours. The time tolerance window for blood samples will be ±1 minute for all samples collected before 8 hours post-dose and ±3 minutes for subsequent samples. Time of blood sampling will be recorded in the CRF.
- Meals as required in section 5.5.1. Time and consumption of meals will be recorded on CRF.
- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.

#### 8.2.3 Period 1/Day 2

- Obtain oral body temperature. The results for each measurement will be recorded in the CRF.
- Collect a blood sample for pharmacokinetic analysis at 24 hours post dosing of Day 1 continuing into Day 2. The time tolerance window for blood sample will be ±3 minutes. Time of blood sampling will be recorded in the CRF.
- Meals as required. Time and consumption of meals will be recorded on CRF.



- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.
- Collect nasal/nasopharyngeal swab sample for COVID-19 test. Date and time of sample collection and test results (positive or negative) will be documented in the CRF.
- After all procedures are completed, subjects are discharged from the clinical site.

#### 8.2.4 Washout Period

• Collect nasal/nasopharyngeal swab sample for COVID-19 test within 24 to 72 hours prior to check-in (Day -1) in Period 2. Date and time of sample collection and test results (positive or negative) will be documented in the CRF.

#### 8.2.5 Period 2/Day -1

After a washout period of at least 7 days after the first dose (Period 1/Day 1), subjects will be admitted to the clinical site the day prior to Day 1 dosing.

The following procedures will be completed following admission to the clinical site:

- Collect nasal/nasopharyngeal swab sample for COVID-19 test. Date and time of sample collection and test results (positive or negative) will be documented in the CRF.
- Brief physical examination including evaluation of general appearance, heart, lung. The results will be recorded in the CRF.
- Obtain oral body temperature. The results for each measurement will be recorded in the CRF.
- Collect urine for drug screening. The results will be recorded in the CRF.
- Collect urine for cotinine screening. The results will be recorded in the CRF.
- Obtain blood for serum  $\beta$ -hCG for all females of childbearing potential. The results will be recorded in the CRF. (note: blood for serum  $\beta$ -hCG can be obtained at admission or in the morning of Day -1)
- Confirm proper contraception is being used and the results will be recorded on the CRF.
- Collect alcohol breath test. Result will be recorded on the CRF.
- Meals as required in section 5.5.1. Time and consumption of meals will be recorded on CRF.



- Subjects will begin fasting at least 10 hours prior to dosing on Day 1.
- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.

## 8.2.6 Period 2/Day 1

**Prior to** dosing, within 1 hour of study drug administration, the following procedures will be completed:

- Obtain seated blood pressure, pulse rate, respiratory rate and oral body temperature. The results for each measurement will be recorded in the CRF.
- Review Inclusion and Exclusion criteria and record in the CRF
- Collect a blood sample for pharmacokinetic analysis. Time of blood sampling will be recorded in the CRF.
- After all pre-dose procedures have been completed, administer the investigational product (see Investigational/Study Products section) and record in the CRF.

After dosing, the following procedures will be completed:

- Collect blood samples for pharmacokinetic analysis at the following time points after dosing on Day 1: 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, and 16 hours. The time tolerance window for blood samples will be ±1 minute for all samples collected before 8 hours post-dose and ±3 minutes for subsequent samples. Time of blood sampling will be recorded in the CRF.
- Meals as required in section 5.5.1. Time and consumption of meals will be recorded on CRF.
- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.

Protocol Number: 218246



## 8.2.7 Period 2/Day 2

- Collect a blood sample for pharmacokinetic analysis at 24 hours post dosing of Day 1 continuing into Day 2. The time tolerance window for blood sample will be ±3 minutes. Time of blood sampling will be recorded in the CRF.
- Meals as required in section 5.5.1. Time and consumption of meals will be recorded on CRF.
- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond
  to a non-leading question such as "How do you feel?" will be assessed and any AEs
  recorded in the CRF.

#### 8.2.8 End of Study

The exit examination procedures will be done before check-out from the clinic, on study Day 2 of Period 2.

- Obtain seated blood pressure, pulse rate, respiratory rate and oral body temperature. The results for each measurement will be recorded in the CRF.
- Conduct brief physical examination. The results will be recorded in the CRF.
- Collect nasal/nasopharyngeal swab sample for COVID-19 test. Date and time of sample collection and test results (positive or negative) will be documented in the CRF.
- Obtain blood and urine samples for safety laboratory tests.
- Collect urine pregnancy test for all females of childbearing potential. The results will be recorded in the CRF.
- Changes in concomitant medication or non-drug treatments/procedures will be documented in the CRF.
- Spontaneous reporting of adverse events and those elicited by asking subjects to respond to a non-leading question such as "How do you feel?" will be assessed and any AEs recorded in the CRF.

## 8.3 Study Conclusion

The Study Conclusion page of the CRF will be completed for all subjects whether they completed all study procedures or if they were discontinued from the study early. If the subject discontinued early, at any point during the study, the primary reason for withdrawal should be recorded on the Study Conclusion page.



If a subject has any clinically significant, study-related abnormalities or AEs at the end of the study, the GSK CH medical monitor (or designated representative) should be notified and, the subject may be asked to remain at the clinical site or be asked to return for a follow-up visit to ensure any issue is resolved or deemed not clinically significant.

## 8.4 Follow-up Visit

The study site may contact a subject to follow up an AE post-study completion/withdrawal and, in some circumstances, request they return to the site for additional follow-up visits (final safety assessments). If needed, additional examinations may be carried out at such visits.

## 9 STUDY ASSESSMENTS

Every effort should be made to ensure that protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances, outside the control of the investigator that may make it unfeasible to complete an assessment. In these cases, the investigator must take all steps necessary to ensure the safety and well-being of the subject. When a protocol-required assessment cannot be performed, the investigator (or designee) will document the reason for the missed assessment as a protocol deviation and any corrective and preventative actions that he or she has taken to ensure that required processes are adhered to as soon as possible. The Sponsor must be informed of any missed assessments in a timely manner.

## 9.1 Screening Assessments

Screening assessments will be performed by appropriately trained staff/clinical examiners at the times, and in the order defined in the Study Procedures section of this protocol

## 9.2 Safety and Other Assessments

The following safety assessments will be performed by appropriately trained staff/clinical examiners, at the times and in the order defined in the Study Procedures section of this protocol.

## 9.2.1 Laboratory Tests

The following laboratory tests/analytical measures will be performed by appropriately trained staff/clinical examiners, at the times and in the order defined in the Study Procedures section of this protocol.

Protocol Number: 218246



#### Table 9-1 Laboratory Tests

| Hematology | Chemistry | Urinalysis | Drug, cotinine, and alcohol screens |
|---|---|---|---|
| Hematocrit Hemoglobin Platelet count RBC count WBC count and differential: Basophils Eosinophils Lymphocytes Monocytes Neutrophils | Albumin ALP ALT AST Calcium Chloride Creatine kinase Creatinine GGT Glucose Phosphorus Potassium Sodium Total bilirubin Total protein Urea (BUN) | Bilirubin Blood (occult) Color and appearance Glucose Ketones Leukocyte esterase Nitrite pH Protein Specific gravity Urobilinogen Microscopic examinationa | Amphetamines /methamphetamines Barbiturates Benzodiazepines Cocaine MDMA Methadone Opiates PCP THC Urine cotinine test Alcohol breath test |
| Serology | Hormone panel - females only | | |
| HBsAg<br>HBcAb (IgG + IgM)<br>HCV Ab<br>HIV antigen/antibody | Serum FSH <sup>b</sup><br>Serum pregnancy test <sup>c</sup><br>Urine pregnancy test <sup>d</sup> | | |

Definitions: RBC= red blood cell; WBC= white blood cells; AST= aspartate transaminase; ALT= alanine transaminase; GGT= gamma-glutamyl transpeptidase; BUN= blood urea nitrogen; MDMA= 3,4- methylenedioxymethamphetamine; PCP= phencyclidine; THC= tetrahydrocannabinol; HBsAg= hepatitis B surface antigen; HBcAb= Hepatitis B core antibody; HCV Ab= hepatitis C virus antibodies; HIV= human immunodeficiency virus; FSH= follicle-stimulating hormone.

Additional laboratory results may be reported on these samples because of the method of analysis or the type of analyzer used by the clinical laboratory; or as derived from calculated values. These additional tests would not require additional collection of blood. Unscheduled

ain the event of abnormal findings

<sup>&</sup>lt;sup>b</sup>FSH done at screening only in females who have been amenorrhoeic for 12 months

<sup>&</sup>lt;sup>c</sup>All female subjects of childbearing potential will be tested for serum human chorionic gonadotropin (hCG) at Day -1 of each period

<sup>&</sup>lt;sup>e</sup>All female subjects of childbearing potential will undergo a urine pregnancy test at Screening and End of Study.



clinical labs may be obtained at any time during the study to assess any perceived safety concerns.

Subjects may undergo random urine drug screening at the discretion of the investigator; the result would be recorded in the CRF. Drug screening conducted prior to dosing must be negative for subjects to receive investigational product.

Any remaining serum/plasma from samples collected for clinical safety labs will be destroyed at the end of the study.

## 9.2.2 Serology

Virus serology will be performed at times specified in the Study Procedures section of this protocol for HIV antigen and antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) (IgG + IgM) and hepatitis C virus antibody (HCV Ab). Serology will be performed by using the same sample drawn for chemistry; therefore, no additional blood needs to be drawn for serology. In case of a positive finding in virus serology screen, the subject must be excluded from trial participation.

#### 9.2.3 Urine drug screen

Urine will be collected at times specified in the Study Procedures section of this protocol. In case of a positive finding for any substance class, the subject must be discontinued from the trial (or excluded from trial participation in case of positive findings at the screening visit).

#### 9.2.4 Alcohol test

An alcohol breath test will be conducted at times specified in the Study Procedures section of this protocol. In case of a positive finding in the alcohol test, the subject must be discontinued from the trial.

#### 9.2.5 Pregnancy Testing

For all female subjects of childbearing potential, a urine pregnancy test, will be performed at screening and end of study and a serum pregnancy test will be performed on Day -1 of each period. Results will be obtained prior to dosing during each period.

The investigator and site personnel will remind subjects at each visit to inform site personnel if their menstrual cycle has changed or if they have any other reason to suspect they may be pregnant (e.g. had unprotected intercourse since the last visit).

A negative pregnancy result is required before the subject may receive the investigational product. Pregnancy tests will also be done whenever one menstrual cycle is missed during the active study period (or when potential pregnancy is otherwise suspected). Pregnancy tests may also be repeated as per request of IRBs/ECs or if required by local regulations.



In the case of a positive confirmed pregnancy, the subject will be withdrawn from administration of investigational product and from the study.

#### 9.2.6 Physical Examinations

Physical examinations may be conducted by a physician, trained physician's assistant, or nurse practitioner as acceptable according to local regulation. A full physical examination will include head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, vascular and neurological systems.

A brief physical examination will be focused on general appearance, the respiratory and cardiovascular systems, as well as towards subject reported symptoms.

Any untoward findings identified on physical exams conducted after the administration of the first dose of investigational product will be captured as an adverse event, if those findings meet the definition of an adverse event.

## 9.2.7 Height and Weight

Height in centimeters (cm) and body weight in kilograms (kg) to the nearest 0.1 kilogram will be measured.

For measuring weight, a scale with appropriate range and resolution is used and must be placed on a stable, flat surface. Subjects must remove shoes, bulky layers of clothing, and jackets so that only light clothing remains. They must also remove the contents of their pockets and remain still until during measurement of weight.

BMI will be calculated in kg/m<sup>2</sup>.

#### 9.2.8 Blood Pressure and Pulse Rate

Additional collection times, or changes to collection times of blood pressure and pulse rate will be permitted, as necessary at the discretion of the investigator, to ensure appropriate collection of safety data.

Seated blood pressure should be measured with the subject's arm supported at the level of the heart and recorded to the nearest mmHg after a minimum 5 minutes of rest. The same arm (preferably the dominant arm) will be used throughout the study.

A calibrated blood pressure cuff of the same proper size will be used to measure blood pressure each time. The use of an automated device for measuring blood pressure and pulse rate is acceptable, although, when done manually, pulse rate will be measured in the brachial/radial artery for at least 30 seconds. When the timing of these measurements coincides with a blood collection, blood pressure and pulse rate should be obtained prior to the nominal time of the blood collection.



#### 9.2.9 Respiratory Rate

Respiratory rate will be measured after approximately 5 minutes rest in seated position by observing and counting the respirations of the subject for 30 seconds and multiplied by 2. When blood pressure is to be taken at the same time, respiration measurement will be done after the 5 minutes of rest and before blood pressure measurement.

#### 9.2.10 Temperature

Body temperature will be measured orally.

#### 9.2.11 COVID-19 Test

Nasal/nasopharyngeal swab will be collected to test for COVID-19 using PCR or antigen test, at times specified in the Study Procedure section. Two consecutive negative tests for active COVID-19 separated by > 24 hours are required for inclusion in the study: one test will be done at screening within 72 hours of admission and one test will be done on Day -1 in Period 1.

For detection of COVID-19, test/s are to be performed as follows:

- During the screening
- At check-in (Day -1 of each period)
- During the washout period
- At discharge from Period 1 and end of study or early discontinuation
- At any time during residential period in study, when subjects report symptoms suggestive of COVID-19

If the first test is > 72 hours prior to unit admission, subjects should be advised to self-quarantine until entrance to the unit while awaiting final testing clearance. Subjects who report symptoms suggestive of COVID-19 while in the research unit should be isolated in the unit or at home and tested for COVID-19 infection using an approved molecular test.

## 9.2.12 Electrocardiogram

A standard 12 lead ECG will be performed at screening. Interpretation of the tracing must be made by a qualified physician or designee and documented on the ECG section of the CRF. Each ECG tracing should be kept in the source documents at the study site. Results or any clinically significant abnormalities should be reported in the CRF. Clinically significant abnormalities should also be recorded on the Adverse Event CRF. Clinically significant findings must be discussed with the GSK CH Clinical Project Lead (CPL) prior to enrolling the subject in the study. Subjects should be in a quiet environment and not speak during the resting period or measurement. Generally, ECGs should not be collected within 3 hours after food or beverage consumption.



## 9.3 Pharmacokinetics (PK)

Twenty-three (23) blood samples will be collected for pharmacokinetic analysis: within 1 hour prior to dosing (pre-dose), and at 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, and 24 hours following dosing in each treatment period. Time zero ("0") as reference for post-dose PK samplings is defined as the time of drug administration. Time zero will be recorded in the CRF. A dead-volume intravenous catheter will be used for blood collection to avoid multiple skin punctures, when appropriate. Otherwise, blood samples will be collected by direct venipuncture.

## 9.3.1 Plasma for analysis of esomeprazole

During all study periods, blood samples (3 mL) to provide a minimum of 1 mL plasma for pharmacokinetic analysis will be collected into appropriately labeled tubes containing  $K_2EDTA$  at times specified in the protocol. The time tolerance window for blood samples will be  $\pm 1$  minute for all samples collected before 8 hours post-dose and  $\pm 3$  minutes for subsequent samples.

The actual times may change but the number of samples will remain the same. All efforts will be made to obtain the pharmacokinetic samples at the exact nominal time relative to dosing.

Samples will be analyzed using a validated analytical method in compliance with applicable standard operating procedures.

The PK samples must be processed and shipped as indicated in the Analytical Methodology Information Sheet (AMIS) to maintain sample integrity. Any deviations from the PK processing steps, including any actions taken, <u>must</u> be documented and reported to the sponsor. On a case-by-case basis, the sponsor may make a determination as to whether sample integrity has been compromised. Any sample deemed outside of established stability, or of questionable integrity, will be considered a protocol deviation.

#### 9.3.2 Shipment of Pharmacokinetic Samples

When applicable, samples will be transported to the assay lab in at least two separate shipments, with each set of aliquots in separate shipments. Once the assay lab confirms receipt of the first shipment, the second set of aliquots may be sent. The samples should be packed on sufficient dry ice to keep them frozen for at least 72 hours.

All PK samples will be stored until they are properly disposed of at the end of its retention period (i.e., until study report is issued), or useful life (i.e., until expiry of stability), upon written request by Sponsor, or upon receipt of a request to destroy the PK samples due to withdrawal of consent. No sample will be retained beyond 2 years from last participant last visit.

Protocol Number: 218246



#### 9.4 Blood Volume

The total blood sampling volume for each subject in this study is approximately 161 mL. The table below reflects approximate sample volumes needed for each measured endpoint. The actual collection times of blood sampling may change, but the total number of PK blood samples will not increase. Additional blood samples may be taken for safety assessments at the discretion of the investigator or GSK CH.

Table 9-2 Blood Volume

| Sample Type | Sample | Number of Sampling Times | | Total Volume | |
|---|---|---|---|---|---|
| | Volume<br>(mL) | Screening | Study Period | End of Study | (mL) |
| Safety Labs | 8 | 1 | | 1 | 16 |
| Serum Pregnancy<br>Test | 3.5 | | 2 | | 7 |
| PK | 3 | | 46 | | 138 |
| TOTAL | | | | | 161 |

This total volume does not include discarded blood from pre-draws used to remove fluid from flushed catheters, if applicable.

#### 10 ADVERSE EVENT AND SERIOUS ADVERSE EVENTS

The investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study product or the study, or that caused the subject to discontinue the study product or study.

## 10.1 Definition of an Adverse Event (AE)

An AE is any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device).

NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study product including any washout or lead-in product (or medical device).

#### **Events Meeting the AE Definition:**

• Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g. ECG, radiological scans, vital sign measurements), including those that worsen from baseline, considered clinically significant in the



medical and scientific judgment of the investigator (i.e., not related to progression of underlying disease).

- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study product administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study product or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

#### **Events NOT meeting the AE definition:**

- Any clinically significant abnormal laboratory findings (if applicable) or other abnormal safety assessments which are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the subject's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the subject's condition.
- Medical or surgical procedure (e.g. endoscopy, appendectomy) is not the AE. The condition that leads to the procedure is an AE (e.g. appendicitis).
- Situations where an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

## 10.2 Definition of a Serious Adverse Event (SAE)

A Serious Adverse Event (SAE) is a particular category of an adverse event where the adverse outcome is serious. If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g. hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

A serious adverse event is any untoward medical occurrence at any dose that:

- Results in death
- Is life-threatening



• The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

## • Requires inpatient hospitalization or prolongation of existing hospitalization

- In general, hospitalization signifies that the subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, or was necessary, the AE should be considered serious
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

## Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g. sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

## • Results in congenital anomaly/birth defect

#### • Other situations:

- Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

**Note:** Classification of an AE as 'serious' is based on the outcome of the event and is a factor in determining reporting requirements.



## 10.3 Time Period and Frequency for Collecting AE and SAE Information

All AEs, and therefore all SAEs will be collected immediately after a subject provides consent to participate in the study by the completion (signature) of the ICF and until 5 days following last administration of the study product.

Medical occurrences that began before obtaining informed consent will be recorded in the Medical History/Current Medical Conditions section of the CRF not the AE section.

All SAEs will be recorded and reported to the sponsor or designee immediately and under no circumstance should this exceed 24 hours. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek AEs or SAEs after the conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event to be reasonably related to the study product or study participation, the investigator must promptly notify the sponsor.

## 10.4 Reporting Procedures

The investigator and any designees are responsible for detecting, documenting and reporting events that meet the definition of an AE and remain responsible for following up on AEs that are serious, considered related to the study product(s), participation in the study, or a study procedure, or that caused the subject to discontinue the study product or study.

Spontaneous reporting of adverse events and those elicited by asking subjects to respond to non-leading such as "How do you feel" will be assessed and any AE's recorded in the CRF and reported appropriately.

The investigator (or medically qualified designee) is to report all directly observed AEs and all AEs spontaneously reported by the study subject. In addition, each study subject will be questioned about AEs.

Each AE is to be assessed to determine if it meets the criteria for a SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate.

When an AE occurs, it is the responsibility of the investigator (or medically qualified designee) to review all documentation (e.g. hospital progress notes, laboratory, and diagnostics reports) related to the event.

The investigator or site staff will then record all relevant information regarding an AE in the CRF and all details relating to an SAE in the paper SAE Form provided.



It is **not** acceptable for the investigator (or medically qualified designee) to send photocopies of the subject's medical records to GSK CH in lieu of completion of the AE CRF page/SAE form

There may be instances when copies of medical records for certain cases are requested by GSK CH. In this instance, all subject identifiers, except for the subject number, will be redacted on the copies of the medical records prior to submission to GSK CH.

The investigator (or medically qualified designee) will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. The diagnosis will then be documented as the AE/SAE where known and not the individual signs/symptoms. (e.g. upper respiratory tract infection, seasonal allergy, etc. instead of runny nose).

AEs elicited by the investigator (or medically qualified designee) in a standard manner at the study visits should also be recorded in the AE section of the CRF and/or using the SAE form (subject to the classification of the AE). Care will be taken not to introduce bias when questioning a subject about any changes in their health. Open-ended and non-leading verbal questioning should be used.

#### 10.4.1 Reporting of an Adverse Event

All AEs will be reported on the AE page of the CRF by the investigator or site staff. It should be noted that the form for collection of SAE information is not the same as the AE CRF. Where the same data are collected, the AE CRF page and the SAE form must be completed in a consistent manner. For example, the same AE term should be used on both. AEs should be reported using concise medical terminology on the CRF as well as on the form for collection of SAE information.

## 10.4.2 Reporting of a Serious Adverse Event

In addition to recording the details of each AE on the AE CRF page, an SAE form should be completed, as fully as possible. Hard copies of the 'paper' SAE form will be provided in the investigator study master file. Original SAE forms will be retained in the investigator study master file.

It is essential to enter the following information:

- Protocol and subject identifiers
- Subject demography
- Description of events, with diagnosis if available
- Investigator opinion of relationship to study product (or study procedure, if appropriate)
- Criterion for seriousness.



The following are desirable and are of particular relevance for investigator and GSK CH assessment of the SAE report:

- Date of onset of AE
- Date AE stopped, if relevant
- Study product start date
- Study product end date if relevant
- Action taken in relation to the study product
- Outcome if known

The SAE form, completed as fully as possible, must be sent to the Case Management Group, Global Clinical Safety and Pharmacovigilance at GSK CH (PPD), with copy to the appropriate GSK CH Study Manager as soon as possible, but not later than 24 hours after study site personnel learn of the event. The GSK CH Study Manager will be responsible for forwarding the SAE form to other GSK CH personnel as appropriate.

## 10.5 Evaluating Adverse Events

#### 10.5.1 Assessment of Intensity

The investigator or medically qualified designee will make an assessment of intensity for each AE reported during the study and will assign it to one of the following categories:

- Mild: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that is sufficiently discomforting to interfere with normal everyday activities
- Severe: An event that prevents normal everyday activities.

NOTE: An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both non-serious AEs and SAEs can be assessed as severe. For example, a headache may be severe (interferes significantly with the subject's usual function) but would not be classified as serious unless it met one of the criteria for SAEs, listed above. An event is defined as 'serious' when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### 10.5.2 Assessment of Causality

The causality assessment is one of the criteria used when determining regulatory reporting requirements.



For each AE (serious and non-serious), the investigator (or medically qualified designee) <u>must</u> provide an assessment of causality on the AE CRF page and the SAE form (subject to the classification of the AE). The investigator will also document in the medical notes that he/she has reviewed the AE and assessed causality, where applicable.

A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out. Generally, the facts (evidence) or arguments to suggest a causal relationship should be provided.

The investigator will use clinical judgment to determine the relationship in the determination of his/her assessment. Alternative causes, such as underlying disease(s), concomitant therapy, other risk factors, and the temporal relationship of the event to the study product will be considered and investigated.

For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.

The investigator's assessment of causality must be provided for all AEs (serious and non-serious); the investigator must record the causal relationship in the CRF, as appropriate, and report such an assessment in accordance with the SAE reporting requirements if applicable.

There may be situations when an SAE has occurred, and the investigator has minimal information to include in the initial report to GSK. However, it is very important that the investigator always make an assessment of causality for every event prior to the initial transmission of the SAE data to GSK CH. The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.

#### 10.6 Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow up with each subject and provide further information on the subject's condition.

All AEs (serious and non-serious) will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up.

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as may be indicated or as requested by GSK CH to elucidate as fully as possible the nature and/or causality of the AE. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

New or updated information will be recorded on the AE CRF page and on the SAE form (subject to the classification of the AE).



The investigator will submit any updated SAE data to GSK CH within 24 hours of receipt of the information.

Investigators are not obliged to actively seek AEs in former subjects. However, if the investigator learns of a SAE, including death, at any time after a subject has been discharged from the study, and considers the event reasonably related to the study product or study participation, the investigator will promptly notify GSK CH by emailing the information to the Case Management Group, Global Clinical Safety and Pharmacovigilance group mailbox at GSK (PPD ) with a copy to the appropriate GSK CH Study Manager. The GSK CH Study Manager will be responsible for forwarding the SAE form to other GSK CH personnel as appropriate.

The investigator will submit any updated SAE data to GSK CH within the designated reporting time frames.

#### 10.7 Withdrawal Due to an Adverse Event

Withdrawal due to AEs should be distinguished from withdrawal due to other causes, according to the definition of an AE noted earlier, and recorded on the appropriate AE CRF page.

When a subject withdraws because of an SAE, the SAE must be reported in accordance with the reporting requirements defined.

## 10.8 Regulatory Reporting Requirements for SAEs

GSK CH has a legal responsibility to notify, as appropriate, the local regulatory authority and other regulatory authorities about the safety of a product under clinical investigation. Prompt notification of SAEs by the investigator to GSK CH is essential so that legal obligations and ethical responsibilities towards the safety of subjects are met.

GSK CH will comply with country specific regulatory requirements relating to safety reporting to the regulatory authority, IRB/EC and investigators.

Both the investigator and the sponsor will comply with all local medical device reporting requirements

Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.

An investigator who receives an investigator safety report describing a SAE or other specific safety information e.g. summary or listing of SAE from the sponsor will review and then file it along with the supporting documentation in the investigator study master file, and will notify the IRB/IEC, if appropriate according to local requirements.



## 10.9 Pregnancy

#### 10.9.1 Time Period for Collecting Pregnancy Information

Pregnancy information will be collected on all pregnancies reported while a female subject is participating in the study from the signing of informed consent until 5 days after last administration of study product.

## 10.9.2 Action to be Taken if Pregnancy Occurs

The investigator will record pregnancy information on the appropriate form, scan and e-mail it to the Case Management Group, Global Clinical Safety and Pharmacovigilance mailbox (PPD ) with a copy to the appropriate GSK CH Study Manager. The GSK CH Study Manager will be responsible for forwarding the pregnancy form to other GSK CH personnel as appropriate. Original pregnancy information forms will be retained in the investigator study master file.

The subject will be followed to determine the outcome of the pregnancy. Information on the status of the mother and infant / neonate (including concomitant medications taken by the mother during the pregnancy) will be forwarded by the investigator the Case Management Group, Global Clinical Safety and Pharmacovigilance group mailbox at GSK (PPD PPD) with a copy to the appropriate GSK CH Study Manager. The GSK CH Study Manager will be responsible for forwarding the pregnancy form to other GSK CH personnel as appropriate. Generally, follow-up will be no longer than 6 to 8 weeks following the estimated delivery date. Any termination of the pregnancy will be reported.

While pregnancy itself is not considered to be an AE, abnormal pregnancy outcomes (e.g. spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are, and should be recorded as an SAE.

Any female subject who becomes pregnant while participating will be withdrawn from the study.

## 10.10 Regulatory Reporting Requirements for Medical Device Incidents

To fulfill regulatory reporting obligations worldwide, the investigator is responsible for the detection and documentation of events meeting the definitions of incident or malfunction that occur during all periods of the study in which the medical device is used.

The investigator will promptly report all incidents occurring with any medical device provided for use in the study in order for the sponsor to fulfill the legal responsibility to notify appropriate regulatory authorities and other entities about certain safety information relating to medical devices being used in clinical studies.



The investigator, or responsible person according to local requirements (e.g. the head of the medical institution), will comply with the applicable local regulatory requirements relating to the reporting of incidents to the IRB/IEC.

## 11 DATA MANAGEMENT

As used in this protocol, the term CRF is understood to refer to either a paper form or an electronic data record or both, depending on the data collection method.

For this study, subject data will be entered into an electronic CRF (eCRF), using a validated system. Data relating to SAEs, pregnancy and incidents will also be collected on paper forms.

The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.

The source documents (e.g. hospital records, clinical and office charts, laboratory notes, memoranda, subject diaries, questionnaires, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files and records kept at the pharmacy, at the laboratory and at the medico-technical departments involved in the clinical study) which contain the source of data recorded in the CRF should be specified. The CRF can be used as a source document at the discretion of data management.

Each subject will be assigned and identified by a unique Screening Subject Number. Any reference made to an individual subject within the study must be done using their unique Screening Subject Number.

## 11.1 Case Report Form

A CRF is a printed, optical, or electronic document designed to record the protocol required information to be reported to the sponsor on each trial subject.

For each subject who has given informed consent/assent the CRF must be completed and signed by the Principal Investigator (or authorized designee) to certify that the data are complete and correct. The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.

Management of clinical data will be performed in accordance with Third Party BDM Vendor applicable standards and data cleaning procedures with oversight by GSK CH to ensure integrity of the data, for example, to remove errors and inconsistencies in the data.

To protect the privacy of subjects, no Personal Information (PI) (including the subject's name or initials or full birth date) is to be recorded in the CRF or as part of the query text.



All CRF pages should be completed during a subject assessment when the CRF has been designated as the source. Data that is sourced elsewhere should be entered into the CRF in an agreed upon timeframe between the Investigator and Sponsor.

GSK CH will obtain and retain all CRFs and associated study data as applicable at the completion of the study.

## 11.2 Data Handling

Documentation of all data management activities should allow step-by-step retrospective assessment of data quality and study performance.

Any changes or corrections to data will be performed in the Electronic Data Capture (EDC) System, and it will include rationale for changes. The EDC system has an audit trail, which will provide a complete record of the changes and corrections endorsed by the Investigator.

Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and any concomitant medications terms (if applicable) using WHO Drug Dictionary (WHO DD).

#### 11.2.1 Data Queries

Programmed edit checks will be generated automatically, as the data are being entered into the system. Reports and listings on the CRF data will also be run, in addition to the queries already programmed and generated by the system, to raise manual queries as needed for site clarification or correction. A query should be issued to update the verbatim towards a codable description.

The study monitor will perform ongoing review of the CRFs in accordance with the monitoring plan, to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

Any queries will be generated in the EDC System to the Investigator or designee, enabling the errors to be addressed in parallel with Data Management review. The study monitor can also run reports and listings on the CRFs, to raise manual queries as needed for site clarification or correction.

#### 11.3 External Data

External Data are subject data obtained externally to the CRF. These data are generated from laboratory instruments, computers or other sources and then transcribed into a file and format agreed upon by GSK CH to identify the subject and time point referenced in the CRF and/or protocol.



An agreed quality control process will be performed against the transcribed data to the source to ensure the accuracy of the transcription. The transcribed data is transmitted in an agreed upon format to GSK CH.

Reconciliation will be performed between the transcribed data and the clinical database to ensure subject and time point referenced in the Clinical Database match before Clinical Database Freeze (locking of the database) can occur.

#### 12 STATISTICAL CONSIDERATIONS AND DATA ANALYSES

## 12.1 Sample Size Determination

A sufficient number of subjects will be screened to randomize approximately 49 to ensure at least 41 evaluable subjects complete the entire study.

According to previous GSK CH study columns, it is estimated a sample of 41 subjects will provide at least 90% power to establish bioequivalence. Considering a drop out discontinuation rate of 15%, approximately 49 subjects will need to be enrolled.

## 12.2 Populations for Analysis

The safety population is defined as all randomized subjects who receive at least one dose of study medication.

The PK population is defined as all randomized subjects who have at least one post-dose PK value, and who have no major protocol deviations concerning pharmacokinetics.

The following PK analysis set is defined to address the PK objectives and further PK considerations within this study:

PK analysis set includes all subjects of the PK population who complete both treatment periods, and for which the relevant PK parameters (at least AUC<sub>0-t</sub> or C<sub>max</sub>) can be derived. Subjects with baseline concentration >5% of the individual C<sub>max</sub> for either period will be excluded from the PK analysis set. This analysis set will be used in summaries, the primary PK analysis, and the secondary PK analysis.

## 12.3 Statistical Analyses

Additional details of the proposed statistical analysis will be documented in the statistical reporting and analysis plan (SAP), which will be written following finalization of the protocol and prior to study unblinding/analysis (as appropriate). This section is a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints.



SAP creation and statistical analysis will be performed by PPD

Pharmacokinetic variables will be calculated by PPD

All concentration and PK data will be listed. This includes any data for subjects who are not included in the analysis (e.g. subjects withdrawn from the study due to adverse events).

## 12.3.1 Primary Analysis(es)

#### Primary Pharmacokinetics Analysis Variables

PK parameters will be derived using the actual sampling times after database lock and unblinding and are defined as follows:

- C<sub>max</sub>: maximum observed post-dose concentration; obtained without interpolation.
- AUC<sub>0-t</sub>: area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule.

#### Statistical Methods:

The bioequivalence between esomeprazole 20 mg delayed-release capsules from CG (test) and esomeprazole 20 mg delayed-release capsules from AZ (Reference) under fasted conditions will be assessed:

- The 90% confidence interval for the ratio of geometric means (test/reference) based on least-squares means from the ANOVA of the ln-transformed AUC<sub>0-t</sub> must be within 0.8 to 1.25; and,
- The ratio of geometric means (test/reference) based on least-squares means from the ANOVA of the In-transformed C<sub>max</sub> must be within 0.8 to 1.25.

A linear mixed effects model will be fit to the log-transformed PK parameters (AUC<sub>0-t</sub> and C<sub>max</sub>), as the dependent variable, and treatment, sequence, and period as fixed effects. Subject nested within sequence will be a random effect. The treatment least-squares means (LSMs), difference between treatment LSMs, and 90% confidence interval (CI) for the difference will be computed. The adjusted mean difference and the 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (test/reference) and 90% CIs for the ratio. If all study subjects are not recruited from the same enrollment pool and the study doses in more than one group, the statistical model may be modified to reflect the multigroup nature of the study. Bioequivalence will be declared for AUC<sub>0-t</sub> if the 90% 2-sided CI for the ratio lies completely within the range of 0.8-1.25 and for C<sub>max</sub> if the point estimate for the ratio lies completely within the range of 0.8-1.25. No further adjustments for multiplicity of the co-primary endpoints are necessary as both endpoints must be met in order to achieve study success.



#### 12.3.2 Secondary Analysis(es)

To further assess the PK profile of esomeprazole the following PK parameters will be derived using actual sampling times:

- AUC<sub>0-inf:</sub> area under the plasma concentration versus time curve calculated from time 0 to infinity AUC<sub>0-inf</sub> = AUC<sub>0-t</sub> + C(t)/ $\lambda_z$  where C(t) is the concentration at the last measurable sampling time point and  $\lambda_z$  is the terminal elimination rate constant.
- %AUC<sub>ex</sub> Percentage of AUC<sub>0-inf</sub> obtained by extrapolation, calculated as  $(1-[AUC_{0-t}/AUC_{0-inf}])\times 100$ .
- $\lambda_z$  terminal elimination rate constant computed as the slope of the regression line of ln (C(t)) on time. The regression should generally involve at least 3 consecutive measurable concentrations that decrease over time.
- t<sub>max</sub>- time of the maximum observed post-dose concentration.
- $t_{1/2}$  elimination half-life computed as  $t_{1/2} = \ln(2)/\lambda_z$ .

The PK parameters (AUC<sub>0-inf</sub>, %AUC<sub>ex</sub>,  $\lambda_z$ ,  $t_{max}$ , and  $t_{1/2}$ ) will be summarized for each treatment using descriptive statistics same as for the primary PK parameters.

#### 12.3.3 Safety Analysis(es)

The assessment of safety will be based on the frequency and severity of treatment emergent AEs (TEAEs) i.e., AEs that are emergent or that worsen after the first study product (test or reference) administration.

The incidence of TEAEs will be summarized by presenting, for each treatment, the number and percentage of subjects having any AE, any AE in each MedDRA System Organ Class (SOC) and having each individual AE. The subset of AEs suspected of a relationship to study drug will be presented in a similar manner. All TEAEs will be also tabulated by severity. Any other information collected (e.g., action taken, duration, outcome) will be listed. AEs will be assigned to the treatment administered immediately prior to the onset. Adverse events due to COVID-19, if any, will be listed and tabulated separately.

Vital signs including temperature will be summarized by time-point and treatment. Summary statistics will include mean, standard deviation, minimum, median, and maximum. No inferential statistics will be presented. Data will be listed with abnormal values flagged.

Medical history and physical examination, as applicable, will be listed with abnormal values flagged.

Laboratory data and ECGs collected at screening and used for inclusion/exclusion criteria will be considered source data, and will not be required to be reported, unless otherwise noted.



#### 12.3.4 Other Analysis(es)

Not applicable.

#### 12.3.5 Exclusion of Data from Analysis

Subjects who deviate from the protocol will be identified and excluded from the pharmacokinetic analyses as agreed by the biostatistician and medical director or designee. Exclusion of subjects with baseline > 5% of the  $C_{max}$  will be determined before database lock and unblinding. Exclusion of any data from the analyses will be determined during a Blind Data Review (BDR) Meeting prior to database lock. Any reasons for exclusion from an analysis population will be listed, if applicable.

#### 12.3.6 Demographic and Baseline Characteristics

Baseline data, relevant screening data, and demographic characteristics will be summarized for all randomized subjects.

## 12.3.7 Study Drug/Product Compliance and Use of Other Therapies

## 12.3.7.1 Study Drug/Product Compliance

The number of subjects exposed to each treatment will be tabulated for the safety population. Treatment deviations for individual subjects will be listed and summarized.

#### 12.3.7.2 Prior and Concomitant Medications

Prior and concomitant medications will be listed for the safety population.

#### 12.3.8 Handling of Dropouts and Missing Data

All existing data for subjects who are dropouts from the study will be included in the pharmacokinetic statistical analysis.

If any concentration data is missing or deviates from the planned time of collection, then the pharmacokineticist may calculate the PK parameters using the available data.

Missing values of  $\lambda_z$  can be estimated from the subject's mean  $\lambda_z$  value from the other treatments. If a  $\lambda_z$  value cannot be calculated from the other treatments, then the  $\lambda_z$  will be obtained from the treatment mean value for subjects with non-missing values of  $\lambda_z$  in the period in which it is not available. This estimated  $\lambda_z$  can be used to calculate other  $\lambda_z$  dependent variables. This  $\lambda_z$  value derivation is only applied for pre-dose concentration adjustments.

For esomeprazole concentration:

• BLOQ values obtained before the first measurable concentration will be imputed as zero.



 BLOQ values obtained after the first measurable concentration will be "Not detectable" (ND), which will be shown as missing (explanations will be specified in the footnote of TFLs).

## 12.3.9 Interim Analysis

No interim analysis is planned for this study

#### 13 STUDY GOVERNANCE CONSIDERATIONS

## 13.1 Quality Control

In accordance with applicable regulations including GCP, and GSK CH procedures, GSK CH or designee (i.e. third-party vendor) monitors will contact the site prior to the start of the study to review with the site staff the protocol, study requirements, and their responsibilities to satisfy regulatory, ethical, and GSK CH requirements.

When reviewing data collection procedures, the discussion will include identification, agreement and documentation of data items for which the CRF will serve as the source document.

GSK CH or designee will monitor the study and site activity to verify that the:

- Data are authentic, accurate, and complete.
- Safety and rights of subjects are being protected.
- Study is conducted in accordance with the currently approved protocol and any other study agreements, GCP, and all applicable regulatory requirements.

The extent and nature of monitoring will be described in a written monitoring plan on file at GSK CH. The investigator (or designee) agrees to allow the monitor direct access to all relevant documents and agrees to co-operate with the monitor to ensure that any problems detected in the course of these monitoring visits are resolved.

## 13.2 Quality Assurance

To ensure compliance with GCP and all applicable regulatory requirements, GSK CH may conduct a quality assurance assessment and/or audit of the site records, and the regulatory agencies may conduct a regulatory inspection at any time during or after completion of the study.

In the event of an assessment, audit or inspection, the investigator (and institution) must agree to grant the advisor(s), auditor(s) and inspector(s) direct access to all relevant documents and to allocate their time and the time of their staff to discuss the conduct of the study, any



findings/relevant issues and to implement any corrective and/or preventative actions to address any findings/issues identified.

The investigator(s) will notify GSK CH or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with GSK CH or its agents to prepare the study site for the inspection and will allow GSK CH or its agent, whenever feasible, to be present during the inspection. The investigator will promptly apply copies of the inspection finding to GSK CH or its agent. Before response submission to the regulatory authority, the investigator will provide GSK CH or its agents with an opportunity to review and comment on responses to any such findings.

The sponsor will be available to help investigators prepare for an inspection.

## 13.3 Regulatory and Ethical Considerations

#### 13.3.1 Institutional Review Board/ Ethics Committee

It is the responsibility of the investigator to have prospective approval of the study protocol, protocol amendments, informed consent documents, investigator brochure/safety statement (including any updates) and other relevant documents, e.g. recruitment advertisements, if applicable, from the IRB/EC. All correspondence with the IRB/EC should be retained in the investigator file. Copies of IRB/EC approvals should be forwarded to GSK CH prior to the initiation of the study, and also when subsequent amendments to the protocol are made.

The only circumstance in which an amendment may be initiated prior to IRB/EC approval is where the change is necessary to eliminate apparent immediate hazards to the subjects. In that event, the investigator must notify the IRB/EC and GSK CH in writing immediately after the implementation.

## 13.3.2 Ethical Conduct of the Study

The study will be conducted in accordance with the protocol and legal and regulatory requirements, as well as the general principles set forth in the International Ethical Guidelines for Biomedical Research Involving Human Subjects (Council for International Organizations of Medical Sciences 2002), International Ethical Guidelines for Health-Related Research Involving Humans (Council for International Organizations of Medical Sciences, 2016), guidelines for GCP (ICH 1996 and revision 2), and the Declaration of Helsinki (World Medical Association 2013).

In addition, the study will be conducted in accordance with the protocol, the ICH guideline on GCP, and applicable local regulatory requirements and laws.



## 13.3.3 Subject Information and Consent

All parties will ensure protection of subject personal data and will not include subject names or other identifiable data in any reports, publications, or other disclosures, except where required by laws.

When study data are compiled for transfer to GSK CH and other authorized parties, subject names, addresses, and other identifiable data will be replaced by numerical codes based on a numbering system provided by GSK CH in order to de-identify study subjects. The use of initials should be avoided.

The study site will maintain a confidential list of subjects who participated in the study, linking each subject's numerical code to his or her actual identity. In case of data transfer, GSK CH will maintain high standards of confidentiality and protection of subjects' personal data consistent with applicable privacy laws.

The informed consent documents must be in compliance with ICH GCP, local regulatory requirements, and legal requirements, including applicable privacy laws.

The informed consent documents used during the informed consent process must be reviewed and approved by the sponsor, approved by the IRB/EC before use, and available for inspection.

The investigator must ensure that each study subject, is fully informed about the nature and objectives of the study and possible risks associated with participation.

The investigator, or a person designated by the investigator, will obtain written informed consent from each subject before any study-specific activity is performed. The investigator will retain the original of each subject's signed informed consent document.

#### 13.3.4 Subject Recruitment

Advertisements approved by IRBs/ECs and investigator databases may be used as recruitment procedures. Use of ethics committee approved, generic, prescreening questionnaire to assess basic subject characteristics to determine general eligibility for this study is allowed. This generic questionnaire may be used by sites as a phone script and/or to review internal databases to identify subjects.

GSK CH will have an opportunity to review and approve the content of any study recruitment materials directed to potential study subjects before such materials are used.

## 13.3.5 Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

Within GSK CH a serious breach is defined as a breach likely to affect to a significant degree the safety and rights of a subject or the reliability and robustness of the data generated in GSK CH-sponsored human subject research studies.



In the event of any prohibition or restriction imposed (i.e., clinical hold) by an applicable competent authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the investigational product, GSK CH should be informed immediately.

In addition, the investigator will inform GSK CH immediately of any urgent safety measures taken by the investigator to protect the study subjects against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP that the investigator becomes aware of.

# 13.4 Posting of Information on Publicly Available Clinical Trial Registers

Study information from this protocol will be posted on publicly available clinical trial registers before enrollment of subjects begins in accordance with applicable GSK CH processes.

GSK intends to make anonymized subject-level data from this trial available to external researchers for scientific analyses or to conduct further research that can help advance medical science or improve patient care. This helps ensure the data provided by trial participants are used to maximum effect in the creation of knowledge and understanding

## 13.5 Provision of Study Results to Investigators

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a GSK CH site or other mutually-agreeable location.

GSK CH will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study subjects, as appropriate.

The procedures and timing for public disclosure of the results summary and for development of a manuscript for publication will be in accordance with GSK CH Policy.

A manuscript will be progressed for publication in the scientific literature if the results provide important scientific or medical knowledge.

#### 13.6 Records Retention

Following closure of the study, the investigator must maintain all site study records (except for those required by local regulations to be maintained elsewhere), in a safe and secure location.

The records (study/ site master file) must be maintained to allow easy and timely retrieval, when needed (e.g. for a GSK CH audit or regulatory inspection) and must be available for review in conjunction with assessment of the facility, supporting systems, and relevant site staff.



Where permitted by local laws/regulations or institutional policy, some or all of these records can be maintained in a format other than hard copy (e.g. microfiche, scanned, electronic); however, caution needs to be exercised before such action is taken.

The investigator must ensure that all reproductions are legible and are a true and accurate copy of the original and meet accessibility and retrieval standards, including re-generating a hard copy, if required. Furthermore, the investigator must ensure there is an acceptable back-up of these reproductions and that an acceptable quality control process exists for making these reproductions.

The investigator must assure that the subject's anonymity will be maintained. On CRFs or other documents submitted to GSK CH, subjects should not be identified by their names or initials, but by an identification code. The investigator should keep a separate log of subjects' codes, names and addresses. Documents not for submission to GSK CH, e.g. subjects' written consent forms, should be maintained by the investigator in strict confidence.

Records and documents, including signed ICF, pertaining to the conduct of this study must be retained by the investigator for 25 years, from the issue of the final Clinical Study Report (CSR) or equivalent summary, unless local regulations or institutional policies require a longer retention period. The minimum retention time will meet the strictest standard applicable to that site for the study, as dictated by any institutional requirements or local laws or regulations, GSK CH standards/procedures, and/or institutional requirements.

No study document should be destroyed without a prior written agreement between GSK CH and the investigator. The investigator must notify GSK CH of any changes in the archival arrangements, including, but not limited to, archival at an off-site facility or transfer of ownership of the records in the event the investigator is no longer associated with the site.

#### 13.7 Conditions for Terminating the Study

Premature termination of this study may occur because of a regulatory authority decision, change in opinion of the IRB/EC, or study product safety problems, or at the discretion of GSK CH. In addition, GSK CH retains the right to discontinue development of esomeprazole formulation at any time.

If a study is prematurely terminated, GSK CH will promptly notify the investigator. After notification, the investigator must promptly contact all participating subjects and should assure appropriate therapy/ follow-up for the subjects. As directed by GSK CH, all study materials must be collected and all CRF's completed to the greatest extent possible. Where required by the applicable regulatory requirements, GSK CH should inform the regulatory authority(ies) and the investigator should promptly inform the IRB/EC and provide the IRB/EC a detailed written explanation of the termination or suspension.



If the IRB/EC terminates or suspends its approval/favorable opinion of a trial, the investigator should promptly notify the GSK CH and provide GSK CH with a detailed written explanation of the termination or suspension.

Upon completion or premature discontinuation of the study, the GSK CH monitor will conduct site closure activities with the investigator or site staff, as appropriate, in accordance with applicable regulations including GCP, and GSK CH Standard Operating Procedures.

#### 14 REFERENCES

- 1. Hatcher RA, Trussell J, Nelson AL, Cates W Jr, Stewart F, Kowal D, editors. Contraceptive Technology. 19th edition. New York: Ardent Media, 2007(b): 28. Available on request
- 2. ICH Topic E6 (R2) Guideline for Good Clinical Practice, Nov 2016.
- 3. World Medical Association Declaration of Helsinki, 64th General Assembly, Fortaleza 2013.
- 4. [Health Canada Guidance document, Comparative Bioavailability Standards: Formulations Used for System Effects July 2018]
- 5. [Health Canada Guidance document, Conduct and Analysis of Comparative Bioavailability Studies September 2018]

Protocol Number: 218246



## 15 APPENDICIES

## 15.1 ABBREVIATIONS

The following is a list of abbreviations that may be used in the protocol.

Table 15-1 Abbreviations

| Abbreviation | Term |
|---|---|
| $\lambda_z$ | terminal elimination rate constant |
| Ab | antibody |
| AE | adverse event |
| Ag | antigen |
| ALP | alkaline phosphatase |
| ALT | alanine transaminase |
| AMIS | analytical methodology information sheet |
| ANOVA | analysis of variance |
| AST | aspartate transaminase |
| AUC <sub>0-t</sub> | area under the concentration-time curve from time 0 to the last measurable sampling time point, t |
| AUC <sub>0-inf</sub> | area under the concentration-time curve from time 0 to infinity |
| %AUC <sub>ex</sub> | percentage of AUC <sub>0-inf</sub> obtained by extrapolation |
| AZ | AstraZeneca |
| BDR | blinded data review |
| BLOQ | below the level of quantification |
| ВМІ | body mass index |
| BP | blood pressure |
| BPM | beats per minute |
| BT | body temperature |
| BUN | blood urea nitrogen |
| CG | Catalent Guayama |
| CI | confidence interval |
| CK | creatine kinase |
| C <sub>max</sub> | peak or maximum observed concentration |
| CPL | clinical project lead |
| CRF | case report form |
| CRO | clinical research organization |
| CSR | clinical study report |
| CTA | clinical trial application |
| CV | coefficient of variation |

Protocol Number: 218246



| Abbreviation | Term |
|---------------------|-----------------------------------------------|
| CYP | cytochrome P450 |
| DIN | drug identification number |
| DM | data management |
| EC | ethics committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EDTA | edetic acid (ethylenediaminetetraacetic acid) |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration (United States) |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GERD | gastroesophageal reflux disease |
| GGT | gamma-glutamyl transpeptidase |
| HBcAb | hepatitis B core antibody |
| HBsAg | hepatitis B surface antigen |
| hCG | human chorionic gonadotropin |
| HCV Ab | hepatitis C virus antibody |
| HIV | human immunodeficiency virus |
| IB | investigator's brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IgG | immunoglobulin G |
| IgM | immunoglobulin M |
| IND | investigational new drug |
| IRB | institutional review board |
| IUD | intrauterine contraceptive device |
| K <sub>2</sub> EDTA | dipotassium ethylene diamine tetraacetic acid |
| LSM | least-squares mean |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MDMA | 3,4- methylenedioxymethamphetamine |
| N/A | not applicable |
| ND | not detectable |
| PCP | phencyclidine |
| PCR | polymerase chain reaction |

Protocol Number: 218246



| Abbreviation | Term |
|------------------|-----------------------------------------------|
| PI | personal information |
| PK | pharmacokinetics |
| PR | pulse rate |
| QTc | corrected QT |
| RBC | red blood cell |
| RR | respiratory rate |
| SAE | serious adverse event |
| SAP | statistical reporting and analysis plan |
| SOC | system organ class |
| SOP | standard operating procedure |
| SRDS | single reference safety document |
| SUSAR | suspected unexpected serious adverse reaction |
| T <sub>1/2</sub> | terminal half-life |
| TBC | to be confirmed |
| TEAE | treatment emergent adverse event |
| TFL | tables, figures and listings |
| THC | tetrahydrocannabinol |
| T <sub>max</sub> | time to reach maximum concentration |
| UK | United Kingdom |
| ULN | upper limit of normal |
| US | United States |
| WBC | white blood cell |
| WHO | World Health Organization |
| WHO DD | WHO drug dictionary |

## Signature Page for $\,218246\ TMF\text{-}218106\ v1.0$

| Reason for signing: Approved | Name: PPD Role: A nature: PPD |
|------------------------------|-------------------------------|
| Reason for signing: Approved | Name: PPD Role: A nature: PPD |
| Reason for signing: Approved | Name: PPD Role: A nature: PPD |

Signature Page for TMF-218106 v1.0